CLINICAL TRIAL: NCT03312907
Title: A Phase 3, Multi-Center, Randomized, Double-Blind, Placebo-Controlled, 104-Week Study to Evaluate the Efficacy and Safety of Belimumab Administered in Combination With Rituximab to Adult Subjects With Systemic Lupus Erythematosus (SLE)
Brief Title: A Study to Evaluate the Efficacy and Safety of Belimumab Administered in Combination With Rituximab to Adult Subjects With Systemic Lupus Erythematosus (SLE) - BLISS-BELIEVE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 205646; 2016-003050-32 (EudraCT Number)
Expanded Access: NCT03125486 (No longer available)
Record Dates: First submitted 2017-10-13; First posted 2017-10-18 (Actual); Results first posted 2022-04-25 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-01

CONDITIONS: Systemic Lupus Erythematosus
Keywords: immunosuppressants; Systemic Lupus Erythematosus Disease Activity Index; Belimumab; Lupus Low Disease Activity State; Systemic Lupus Erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — belimumab; Rituximab; Standard of Care

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Belimumab + Placebo (Placebo Comparator): Eligible subjects will receive Belimumab 200 milligrams (mg) to be administered subcutaneously (SC) on Day 1 and then weekly (i.e., every 7 days) through Week 52. Subjects will also receive rituximab-placebo to be administered by intravenous (IV) infusions at Weeks 4 and 6 in double blind manner. Subjects will receive standard therapy excluding Immunosuppressants and including anti-malarials, non-steroidal anti-inflammatory drugs (NSAIDs), and/or corticosteroids tapered down to prednisone equivalent of less than or equal to (<=) 5 mg/day until Week 104. Subjects will not receive treatment after 52 weeks and will be in observation until Week 104.
  Interventions: Drug: Belimumab; Drug: Rituximab-placebo; Drug: Standard therapy (Excluding Immunosuppressants); Drug: Steroid Taper
- Belimumab + Rituximab (Experimental): Eligible subjects will receive Belimumab 200 mg to be administered SC on Day 1 and then weekly (i.e., every 7 days) through Week 52. Subjects will also receive rituximab 1000 mg to be administered by IV infusions at Weeks 4 and 6 in double blind manner. Subjects will receive standard therapy excluding Immunosuppressants and including anti-malarials, NSAIDs, and/or corticosteroids tapered down to prednisone equivalent of <= 5 mg/day until Week 104. Subjects will not receive treatment after 52 weeks and will be in observation until Week 104.
  Interventions: Drug: Belimumab; Drug: Rituximab; Drug: Standard therapy (Excluding Immunosuppressants); Drug: Steroid Taper
- Belimumab + Standard therapy (Other): Eligible subjects will receive open-label Belimumab 200 mg administered SC on Day 1 and then weekly (i.e., every 7 days) until Week 104. Subjects will also receive standard therapy including immunosuppressant, anti-malarials, NSAIDs, and/or corticosteroids tapered down to prednisone equivalent of <= 5 mg/day until Week 104.
  Interventions: Drug: Belimumab; Drug: Standard therapy (Including Immunosuppressants); Drug: Steroid Taper

INTERVENTIONS:
Drug: Belimumab — Belimumab will be administered as SC injection once weekly via autoinjector in thigh or abdomen
Drug: Rituximab — Rituximab will be administered as IV infusion of 1000mg at Week 4 and Week 6
  Arms: Belimumab + Rituximab
Drug: Rituximab-placebo — Saline will be administered as IV infusions at Week 4 and Week 6
  Arms: Belimumab + Placebo
Drug: Standard therapy (Including Immunosuppressants) — Standard therapy will contain stable SLE medications including immunosuppressant to be administered from baseline through Week 104.
  Arms: Belimumab + Standard therapy
Drug: Standard therapy (Excluding Immunosuppressants) — Standard therapy excluding Immunosuppressant will contain anti-malarials, NSAIDs, and/or corticosteroids with prednisone dose equivalent to <= 5 mg/day will administered through Week 104.
  Arms: Belimumab + Placebo; Belimumab + Rituximab
Drug: Steroid Taper — Steroid taper will include prednisone doses equivalent to =< 5 mg/day in all Arms through Week 104.

SUMMARY:
The purpose of this study is to assess whether co-administration of belimumab and a single cycle of rituximab will optimize treatment with belimumab, which will result in improvements of clinical status with a favorable safety profile, by comparing subjects randomized to belimumab plus rituximab versus belimumab plus rituximab-placebo. Approximately 292 subjects will be randomized in a 1:2:1 ratio to 1 of 3 treatment arms; belimumab plus rituximab-placebo (Arm A, control), belimumab plus rituximab (Arm B, combination), or belimumab plus standard therapy (Arm C, reference). Belimumab will be administered as subcutaneous (SC) and rituximab-placebo or rituximab will be administered by intravenous (IV) infusions. The total duration of the study is for 104 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be >=18 years of age at the time of signing the informed consent.
* Subjects who have clinical diagnosis of SLE based on 4 or more of the 11 American College of Rheumatology (ACR) criteria.
* Subjects who have a screening SLEDAI-2K score >=6 (This refers to the total score. Serological activity, i.e., anti-double stranded deoxyribonucleic acid [dsDNA]) positivity and/or hypocomplementemia is not required to be present in SLEDAI-2K assessment, but are scored if present).
* Subjects who have unequivocally positive autoantibody test results defined as an anti-nuclear (ANA) titer >=1:80 and/or a positive anti-dsDNA (>=30 International Units per milliliter [IU/mL]) serum antibody test from 2 independent time points as follows: Positive test results from 2 independent time points within the study screening period. Screening results must be based on the study's central laboratory results. Or, one positive historical test result and 1 positive test result during the screening period.
* Subjects who are on a stable SLE treatment regimen consisting of any of these medications (alone or in combination) for a period of at least 30 days prior to Day 1 (i.e. day of first dose of study treatment) with the exception that switching one agent for another of the same class for tolerability or availability reasons, which will be allowed within 30 days of Day 1: Corticosteroids (prednisone or prednisone equivalent); For those subjects on alternating daily doses of steroids, use the average of 2 daily doses to calculate the average daily steroid dose; Any immunosuppressant or immunomodulatory agents including methotrexate, azathioprine, leflunomide, mycophenolate (including mycophenolate mofetil, mycophenolate mofetil hydrochloride, and mycophenolate sodium), calcineurin inhibitors (example [e.g.] tacrolimus, cyclosporine), sirolimus, oral cyclophosphamide, 6-mercaptopurine, mizoribine, or thalidomide; Anti-malarials (e.g., hydroxychloroquine, chloroquine, quinacrine); Non steroidal anti-inflammatory drugs (NSAIDs).
* Male and/or female. A female subject is eligible to participate if she is not pregnant not breastfeeding, and at least one of the these conditions applies: Not a woman of childbearing potential (WOCBP) or A WOCBP who agrees to follow the contraceptive guidance during the treatment period and for at least 16 weeks after the last dose of belimumab, or at least 12 months after the last dose of rituximab or rituximab-placebo.
* Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.

Exclusion Criteria:

* Symptomatic herpes zoster within 3 months prior to screening.
* Evidence of active or latent tuberculosis (TB). Documentation may include medical history and examination, chest X-rays (posterior, anterior, and lateral), and TB testing: either a positive tuberculin skin test (TST; defined as a skin induration ≥5 mm at 48 to 72 hours, regardless of Baccillus Calmette-Guerin (BCG) or other vaccination history) or a positive (not indeterminate) QuantiFERON-TB Gold Plus test.
* Significant allergies to humanized monoclonal antibodies.
* History of hypersensitivity to belimumab and/or rituximab or known to have titers of human anti-mouse antibody or history of hypersensitivity reactions when treated with other diagnostic or therapeutic monoclonal antibodies.
* Lymphoma, leukemia, or any malignancy within the past 5 years (yrs) except for basal cell or squamous epithelial carcinomas of the skin that have been resected with no evidence of metastatic disease for 3 yrs.
* Alanine transferase (ALT) greater than 2 times upper limit of normal (ULN).
* Bilirubin greater than 1.5 times ULN (isolated bilirubin greater than 1.5 times ULN is acceptable if bilirubin is fractionated and direct bilirubin less than 35%).
* Immunoglobulin A (IgA) deficiency (IgA level less than 10 milligram per deciliter [mg/dL]).
* Immunoglobulin G (IgG) less than 250 mg/dL. For Germany only, IgG less than 400mg/dL.
* Neutrophils less than 1.5 times 10^9.
* Current unstable liver or biliary disease per investigator assessment defined by the presence of ascites, encephalopathy, coagulopathy, hypoalbuminemia, esophageal or gastric varices, persistent jaundice, or cirrhosis.
* Severe heart failure (New York Heart Association Class IV) or other severe, uncontrolled cardiac disease.
* QT interval corrected (QTc) greater than 450 millisecond (msec) or QTc greater than 480 msec in subjects with bundle branch block.
* Subjects who have a history of a major organ transplant (e.g., heart, lung, kidney, liver) or hematopoietic stem cell/marrow transplant.
* Subjects who have clinical evidence of significant unstable or uncontrolled acute or chronic diseases not due to SLE (i.e., cardiovascular, pulmonary, hematologic, gastrointestinal, hepatic, renal, neurological, psychiatric, malignancy, or infectious diseases) which, in the opinion of the principal investigator, could confound the results of the study or put the subject at undue risk.
* Subjects who have an acute or chronic infection requiring management as : Currently on any suppressive therapy for a chronic infection such as pneumocystis, cytomegalovirus, herpes simplex virus, herpes zoster, or atypical mycobacteria); Hospitalization for treatment of infection within 60 days of Day 1; subjects who had infection requiring treatment with parenteral (IV or intramuscular [IM]) antibiotics (antibacterials, antivirals, anti-fungals, or anti-parasitic agents) within 60 days of Day 1. Prophylactic anti-infective treatment is allowed.
* Subjects who have severe lupus kidney disease (defined by proteinuria greater than 6 gram (g)/24 hours or equivalent using spot urine protein to creatinine ratio, or serum creatinine greater than 2.5 mg/dL), or have severe active nephritis requiring induction therapy not permitted by protocol (e.g., IV cyclophosphamide), or have required hemodialysis or high dose prednisone or equivalent (greater than 100 mg/day) within 90 days of Day 1.
* Subjects who have severe active central nervous system (CNS) lupus (including seizures, psychosis, organic brain syndrome, cerebrovascular accident [CVA], cerebritis, or CNS vasculitis) requiring therapeutic intervention within 60 days of Day 1.
* Subjects who have a planned surgical procedure, laboratory abnormality, or condition (e.g., poor venous access) that, in the opinion of the principal investigator, makes the subject unsuitable for the study.
* Subjects who have evidence of serious suicide risk, including any history of suicidal behavior in the last 6 months and/or any suicidal ideation of type 4 or 5 on the Columbia-Suicide Severity Rating Scale (C-SSRS) in the last 2 months or who, in the investigator's opinion, pose a significant suicide risk.
* Subjects who have a history of an anaphylaxis reaction to parenteral administration of contrast agents, human or murine proteins, or monoclonal antibodies.
* Subjects who have received live vaccine(s) within 1 month prior to screening, or plans to receive such vaccines during the screening period or during the study.
* Subjects who have received any of the these prior/concomitant therapy within 364 days of Day 1: Belimumab; Rituximab; Abatacept; Any B cell targeted therapy (anti-cluster of differentiation-20 [CD] agents other than rituximab, anti CD22 [epratuzumab], anti-CD52 [alemtuzumab], BLyS-receptor fusion protein [BR3], Trans-membrane activator and calcium-modulator and cytophilin ligand interactor [TACI] Fc, anti B-cell activating factor [BAFF] (LY2127399), anti-Interferon alpha agents or anti-BLyS other than belimumab); A biologic investigational agent other than B cell targeted therapy (e.g., abetimus sodium, anti CD40L antibody [BG9588/ IDEC 1311]). (Investigational agent applies to any drug not approved for sale in the country in which it is being used).
* Subjects who have required 3 or more courses of systemic corticosteroids within 364 days of Day 1. (Topical or inhaled steroids are permitted).
* Subjects who have received any of these within 90 days of Day 1: Anti- Tumor Necrosis Factor (Anti-TNF) therapy (e.g., adalimumab, etanercept, infliximab); Interleukin-1 receptor antagonist (anakinra); Intravenous immunoglobulin (IVIG); High dose prednisone or equivalent (greater than 100 mg/day); Plasmapheresis.
* Subjects who have received any of the these within 60 days of Day 1: A non-biologic investigational agent (Investigational agent applies to any drug not approved for sale in the country in which it is being used); IV cyclophosphamide and, for Germany only, oral cyclophosphamide; Any steroid injection (e.g., intramuscular [IM], intraarticular, or IV).
* Positive immunodeficiency virus (HIV) antibody test.
* Positive serology for Hepatitis B (HB), defined as HB surface antigen positive (HBsAg+) OR HB core antibody positive (HBcAb+).
* Positive Hepatitis C (HCV) antibody test.
* Subjects who have current drug or alcohol dependence, or a history of drug or alcohol abuse or dependence within 364 days prior to Day 1.
* Sensitivity to any of the study treatments, or components thereof, or drug or other allergy that, in the opinion of the investigator, contraindicates participation in the study.
* Unable to administer study treatment (belimumab) by SC injection and has no other reliable resource to administer the injection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 292 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2020-05-29 (Actual); Study Completion 2021-07-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (73):
- United States (25):
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, La Mesa, California
  - GSK Investigational Site, San Leandro, California
  - GSK Investigational Site, Upland, California
  - GSK Investigational Site, Denver, Colorado
  - GSK Investigational Site, Aventura, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, Tamarac, Florida
  - GSK Investigational Site, Tampa, Florida
  - GSK Investigational Site, Ann Arbor, Michigan
  - GSK Investigational Site, Brighton, Michigan
  - GSK Investigational Site, Lansing, Michigan
  - GSK Investigational Site, Las Cruces, New Mexico
  - GSK Investigational Site, Manhasset, New York
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Charlotte, North Carolina
  - GSK Investigational Site, Vandalia, Ohio
  - GSK Investigational Site, Oklahoma City, Oklahoma
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, Summerville, South Carolina
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, League City, Texas
  - GSK Investigational Site, Spokane, Washington
  - GSK Investigational Site, Glendale, Wisconsin
- Argentina (3):
  - GSK Investigational Site, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - GSK Investigational Site, La Plata, Buenos Aires
  - GSK Investigational Site, San Miguel de Tucumán, Tucumán Province
- Brazil (4):
  - GSK Investigational Site, Salvador, Estado de Bahia
  - GSK Investigational Site, Cuiabá, Mato Grosso
  - GSK Investigational Site, Juiz de Fora, Minas Gerais
  - GSK Investigational Site, São José do Rio Preto, São Paulo
- Canada (4):
  - GSK Investigational Site, Hamilton, Ontario
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Trois-Rivières, Quebec
  - GSK Investigational Site, Saskatoon, Saskatchewan
- France (5):
  - GSK Investigational Site, Brest
  - GSK Investigational Site, Lille
  - GSK Investigational Site, Paris
  - GSK Investigational Site, Pessac
  - GSK Investigational Site, Strasbourg
- Germany (3):
  - GSK Investigational Site, Hanover, Lower Saxony
  - GSK Investigational Site, Kiel, Schleswig-Holstein
  - GSK Investigational Site, Frankfurt
- Mexico (2):
  - GSK Investigational Site, Zapopan, Jalisco
  - GSK Investigational Site, Mérida, Yucatán
- Netherlands (5):
  - GSK Investigational Site, Amersfoort
  - GSK Investigational Site, Groningen
  - GSK Investigational Site, Leiden
  - GSK Investigational Site, The Hague
  - GSK Investigational Site, Utrecht
- Russia (12):
  - GSK Investigational Site, Chelyabinsk
  - GSK Investigational Site, Kazan'
  - GSK Investigational Site, Kemerovo
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Novosibirsk
  - GSK Investigational Site, Omsk
  - GSK Investigational Site, Petrozavodsk
  - GSK Investigational Site, Ryazan
  - GSK Investigational Site, Saint Petersburg
  - GSK Investigational Site, Ufa
  - GSK Investigational Site, Ulyanovsk
  - GSK Investigational Site, Yaroslavl
- South Korea (5):
  - GSK Investigational Site, Daegu
  - GSK Investigational Site, Gwangju
  - GSK Investigational Site, Incheon
  - GSK Investigational Site, Seoul
  - GSK Investigational Site, Suwon
- Spain (5):
  - GSK Investigational Site, Badalona
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Valencia
  - GSK Investigational Site, Valladolid
  - GSK Investigational Site, Vigo (Pontevedra)

IPD SHARING:
Plan to Share IPD: Yes
GSK will assess requests from qualified researchers for anonymized individual patient-level data (IPD) and related study documents. Data sharing is subject to certain criteria, conditions, and exceptions. For further information, refer to https://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD is made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or terminated asset(s) across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf

REFERENCES:
- [Background] Aranow C, Allaart CF, Amoura Z, Bruce IN, Cagnoli PC, Chatham WW, Clark KL, Furie R, Groark J, Urowitz MB, van Vollenhoven R, Daniels M, Fox NL, Gregan YI, Henderson RB, van Maurik A, Ocran-Appiah JC, Oldham M, Roth DA, Shanahan D, Tak PP, Teng YO. Efficacy and safety of sequential therapy with subcutaneous belimumab and one cycle of rituximab in patients with systemic lupus erythematosus: the phase 3, randomised, placebo-controlled BLISS-BELIEVE study. Ann Rheum Dis. 2024 Oct 21;83(11):1502-1512. doi: 10.1136/ard-2024-225686. PMID 39159997
- [Derived] Arends EJ, Zlei M, Tipton CM, Cotic J, Osmani Z, de Bie FJ, Kamerling SWA, van Maurik A, Dimelow R, Gregan YI, Fox NL, Rabelink TJ, Roth DA, Sanz I, van Dongen JJM, van Kooten C, Teng YKO. Disruption of memory B-cell trafficking by belimumab in patients with systemic lupus erythematosus. Rheumatology (Oxford). 2024 Sep 1;63(9):2387-2398. doi: 10.1093/rheumatology/keae286. PMID 38775637
- [Derived] Hannon CW, McCourt C, Lima HC, Chen S, Bennett C. Interventions for cutaneous disease in systemic lupus erythematosus. Cochrane Database Syst Rev. 2021 Mar 9;3(3):CD007478. doi: 10.1002/14651858.CD007478.pub2. PMID 33687069
- [Derived] Teng YKO, Bruce IN, Diamond B, Furie RA, van Vollenhoven RF, Gordon D, Groark J, Henderson RB, Oldham M, Tak PP. Phase III, multicentre, randomised, double-blind, placebo-controlled, 104-week study of subcutaneous belimumab administered in combination with rituximab in adults with systemic lupus erythematosus (SLE): BLISS-BELIEVE study protocol. BMJ Open. 2019 Mar 20;9(3):e025687. doi: 10.1136/bmjopen-2018-025687. PMID 30898822
- [Derived] Parodis I, Lopez Benavides AH, Zickert A, Pettersson S, Moller S, Welin Henriksson E, Voss A, Gunnarsson I. The Impact of Belimumab and Rituximab on Health-Related Quality of Life in Patients With Systemic Lupus Erythematosus. Arthritis Care Res (Hoboken). 2019 Jun;71(6):811-821. doi: 10.1002/acr.23718. PMID 30055091

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a multicenter study conducted at 71 centers in 11 countries. This was a randomized, placebo-controlled, parallel study where participants received treatment in any one of the treatment arms.
Pre-assignment Details: A total of 396 participants were screened, of which 104 were screen failures. A total of 292 participants were enrolled in the study (Intent-to-Treat Population: It comprised of all randomized participants who received at least one dose of study treatment [Belimumab or Rituximab or Placebo]).
Groups:
- Belimumab + Placebo: Participants received Belimumab 200 milligrams (mg) administered subcutaneously (SC) on Day 1 and then weekly (i.e., every 7 days) through Week 52. Participants also received rituximab-placebo administered by intravenous (IV) infusions at Weeks 4 and 6 in double blind manner. Participants received standard therapy excluding Immunosuppressants and including anti-malarials, non-steroidal anti-inflammatory drugs (NSAIDs), and/or corticosteroids tapered down to prednisone equivalent of less than or equal to (<=) 5 mg/day until Week 104. Participants did not receive treatment after 52 weeks and were in observation until Week 104.
- Belimumab + Rituximab: Participants received Belimumab 200 mg administered SC on Day 1 and then weekly (i.e., every 7 days) through Week 52. Participants also received rituximab 1000 mg administered by IV infusions at Weeks 4 and 6 in double blind manner. Participants received standard therapy excluding Immunosuppressants and including anti-malarials, NSAIDs, and/or corticosteroids tapered down to prednisone equivalent of <= 5 mg/day until Week 104. Participants did not receive treatment after 52 weeks and were in observation until Week 104.
- Belimumab + Standard Therapy: Participants received open-label Belimumab 200 mg administered SC on Day 1 and then weekly (i.e., every 7 days) until Week 104. Participants also received standard therapy including immunosuppressant, anti-malarials, NSAIDs, and/or corticosteroids tapered down to prednisone equivalent of <= 5 mg/day until Week 104.
Period: Overall Study
Arm/Group | Belimumab + Placebo | Belimumab + Rituximab | Belimumab + Standard Therapy
Started | 72 | 144 | 76
Completed | 55 | 114 | 57
Not Completed | 17 | 30 | 19
Not completed — Adverse Event | 1 | 6 | 1
Not completed — Protocol Violation | 2 | 3 | 4
Not completed — Lost to Follow-up | 2 | 3 | 2
Not completed — Physician Decision | 3 | 4 | 2
Not completed — Withdrawal by Subject | 9 | 14 | 10

BASELINE CHARACTERISTICS:
Population: Baseline characteristics were presented for Intent-to-Treat Population.
Groups:
- Total: Total of all reporting groups
Arm/Group | Belimumab + Placebo | Belimumab + Rituximab | Belimumab + Standard Therapy | Total
Number analyzed (Participants) | 72 | 144 | 76 | 292
Age, Continuous [Mean (Standard Deviation); unit: Years] | 40.6 (12.58) | 40.1 (11.45) | 41.0 (12.75) | 40.5 (12.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 66 | 129 | 73 | 268
  Male | 6 | 15 | 3 | 24
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White -Arabic/North African Heritage | 0 | 1 | 1 | 2
  White-White/Caucasian/European Heritage | 39 | 100 | 47 | 186
  Asian - Central/South Asian Heritage | 0 | 1 | 1 | 2
  Asian - East Asian Heritage | 7 | 14 | 10 | 31
  Asian - South East Asian Heritage | 3 | 2 | 1 | 6
  African American/African Heritage | 21 | 22 | 13 | 56
  American Indian or Alaskan Native | 1 | 3 | 3 | 7
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a State of Disease Control at Week 52
Description: Percentage of participants with a state of disease control (Independent blinded assessor [IBA]) was defined as the percentage of participants with a Systemic Lupus Erythematosus Disease Activity Index 2000(SLEDAI-2K)score less than or equal to(<=)2 achieved without immunosuppressants and with corticosteroids at a prednisone equivalent dose of <=5 mg/day at Week 52. SLEDAI-2K was a weighted, cumulative index for measuring systemic lupus erythematosus (SLE) disease activity in previous 10 days,consisting 24 individual items in which signs and symptoms, laboratory tests and physician's assessment for each item within each of 9 organ systems were given a weighted score(1 to 8 with higher score indicating increased activity)and summed if present at the time of visit or in preceding 10 days. The SLEDAI-2K score was sum of all 24 individual items from the SLEDAI-2K, ranges from 0(no symptoms) to 105(presence of all defined symptoms) with higher scores representing increased disease activity.
Time Frame: Week 52
Population: Modified Intent-to-Treat (MITT) Population comprised of all randomized participants who received at least one dose of study treatment (Belimumab or Rituximab or Placebo) and excluding participants from Arm 3 (Belimumab + Standard therapy) who were randomized prior to 07-Sep-2018.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Belimumab + Placebo | Belimumab + Rituximab | Belimumab + Standard Therapy
Number analyzed (Participants) | 72 | 144 | 47
Percentage of participants | 16.7 [8.1 to 25.3] | 19.4 [13.0 to 25.9] | 25.5 [13.1 to 38.0]
Statistical Analysis 1: Comparison: Belimumab + Placebo vs Belimumab + Rituximab; Test type: Other; p = 0.5342, Regression, Logistic; Odds Ratio (OR) = 1.27, 95% CI 2-sided [0.60 to 2.71] — Odds ratio was calculated using logistic regression model with covariates: Baseline SLEDAI-2K, Baseline immunosuppressant, Baseline prednisone equivalent dose. Belimumab + Standard therapy arm was excluded from model
Statistical Analysis 2: Comparison: Belimumab + Rituximab vs Belimumab + Standard Therapy; Test type: Other; Odds Ratio (OR) = 0.71, 95% CI 2-sided [0.32 to 1.54] — Odds ratio was calculated using logistic regression model with covariates: Baseline SLEDAI-2K, Baseline immunosuppressant, and Baseline prednisone equivalent dose. Belimumab + Placebo arm excluded from model

2. Secondary Outcome: Percentage of Participants With a State of Clinical Remission at Week 64
Description: Percentage of participants with a state of clinical remission (IBA) was defined as percentage of participants with a clinical SLEDAI-2K score =0 (does not include anti-double stranded deoxyribonucleic [dsDNA] and complement activity scores), achieved without immunosuppressants and with corticosteroids at a prednisone equivalent dose of 0 mg/day at Week 64. SLEDAI-2K was a weighted, cumulative index for measuring SLE disease activity in previous 10 days, consisting 24 individual items in which signs and symptoms, laboratory tests, and physician's assessment for each item within each of 9 organ systems were given a weighted score (1 to 8 with higher score indicating increased activity) and summed if present at the time of the visit or in the preceding 10 days. The clinical SLEDAI-2K score was sum of 22 out of all 24 individual items from the SLEDAI-2K and ranges from 0 (no symptoms) to 101 (presence of all defined symptoms) with higher scores representing increased disease activity.
Time Frame: Week 64
Population: Modified Intent-to-Treat (MITT) Population
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Belimumab + Placebo | Belimumab + Rituximab | Belimumab + Standard Therapy
Number analyzed (Participants) | 72 | 144 | 47
Percentage of participants | 5.6 [0.3 to 10.8] | 6.3 [2.3 to 10.2] | 10.6 [1.8 to 19.5]
Statistical Analysis 1: Comparison: Belimumab + Placebo vs Belimumab + Rituximab; Test type: Other; p = 0.8582, Regression, Logistic; Odds Ratio (OR) = 1.12, 95% CI 2-sided [0.33 to 3.78] — Odds ratio was calculated using logistic regression model with covariates: Baseline SLEDAI-2K, Baseline immunosuppressant, Baseline prednisone equivalent dose and treatment group. Belimumab + Standard therapy arm was excluded from model
Statistical Analysis 2: Comparison: Belimumab + Rituximab vs Belimumab + Standard Therapy; Test type: Other; Odds Ratio (OR) = 0.53, 95% CI 2-sided [0.17 to 1.70] — Odds ratio was calculated using logistic regression model with covariates: Baseline SLEDAI-2K, Baseline immunosuppressant, Baseline prednisone equivalent dose and treatment group. Belimumab + Placebo arm was excluded from model

3. Secondary Outcome: Percentage of Participants With a State of Disease Control at Week 104
Description: Percentage of participants with a state of disease control (IBA) was defined as the percentage of participants with a SLEDAI-2K score <=2, achieved without immunosuppressants and with corticosteroids at a prednisone equivalent dose of <=5 mg/day at Week 104. SLEDAI-2K was a weighted, cumulative index for measuring SLE disease activity in previous 10 days which consisted of 24 individual items in which signs and symptoms, laboratory tests, and physician's assessment for each item within each of 9 organ systems were given a weighted score (1 to 8 with higher score indicating increased activity) and summed if present at the time of the visit or in the preceding 10 days. The SLEDAI-2K score was the sum of all 24 individual items from the SLEDAI-2K which ranges from 0 (no symptoms) to 105 (presence of all defined symptoms) with higher scores representing increased disease activity.
Time Frame: Week 104
Population: Modified Intent-to-Treat (MITT) Population
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Belimumab + Placebo | Belimumab + Rituximab | Belimumab + Standard Therapy
Number analyzed (Participants) | 72 | 144 | 47
Percentage of participants | 6.9 [1.1 to 12.8] | 11.1 [6.0 to 16.2] | 21.3 [9.6 to 33.0]
Statistical Analysis 1: Comparison: Belimumab + Placebo vs Belimumab + Rituximab; Test type: Other; p = 0.3613, Regression, Logistic; Odds Ratio (OR) = 1.64, 95% CI 2-sided [0.57 to 4.72] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Belimumab + Rituximab vs Belimumab + Standard Therapy; Test type: Other; Odds Ratio (OR) = 0.45, 95% CI 2-sided [0.19 to 1.09] — Odds ratio was calculated using logistic regression model with covariates: Baseline SLEDAI-2K, Baseline immunosuppressant, Baseline prednisone equivalent dose and treatment group. Belimumab + Placebo arm excluded from model

4. Secondary Outcome: Percentage of Participants With a State of Disease Control by Visits
Description: Percentage of participants with a state of disease control (IBA) was defined as the percentage of participants with a SLEDAI-2K score <=2, achieved without immunosuppressants and with corticosteroids at a prednisone equivalent dose of <=5 mg/day. SLEDAI-2K was a weighted, cumulative index for measuring SLE disease activity in previous 10 days which consisted of 24 individual items in which signs and symptoms, laboratory tests, and physician's assessment for each item within each of 9 organ systems were given a weighted score (1 to 8 with higher score indicating increased activity) and summed if present at the time of the visit or in the preceding 10 days. The SLEDAI-2K score was the sum of all 24 individual items from the SLEDAI-2K which ranges from 0 (no symptoms) to 105 (presence of all defined symptoms) with higher scores representing increased disease activity.
Time Frame: Weeks 12, 26, 40, 52, 64, 80 and 104
Population: Modified Intent-to-Treat (MITT) Population
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Belimumab + Placebo | Belimumab + Rituximab | Belimumab + Standard Therapy
Number analyzed (Participants) | 72 | 144 | 47
Percentage of participants
  Week 12 | 8.3 [1.9 to 14.7] | 12.5 [7.1 to 17.9] | 21.3 [9.6 to 33.0]
  Week 26 | 16.7 [8.1 to 25.3] | 21.5 [14.8 to 28.2] | 25.5 [13.1 to 38.0]
  Week 40 | 13.9 [5.9 to 21.9] | 20.8 [14.2 to 27.5] | 23.4 [11.3 to 35.5]
  Week 52 | 16.7 [8.1 to 25.3] | 19.4 [13.0 to 25.9] | 25.5 [13.1 to 38.0]
  Week 64 | 11.1 [3.9 to 18.4] | 18.1 [11.8 to 24.3] | 25.5 [13.1 to 38.0]
  Week 80 | 6.9 [1.1 to 12.8] | 13.2 [7.7 to 18.7] | 27.7 [14.9 to 40.4]
  Week 104 | 6.9 [1.1 to 12.8] | 11.1 [6.0 to 16.2] | 21.3 [9.6 to 33.0]

5. Secondary Outcome: Percentage of Participants With a State of Clinical Remission by Visits
Description: Percentage of participants with a state of clinical remission (IBA) was defined as percentage of participants with a clinical SLEDAI-2K score =0 (does not include anti-dsDNA and complement activity scores), achieved without immunosuppressants and with corticosteroids at a prednisone equivalent dose of 0 mg/day. SLEDAI-2K was a weighted, cumulative index for measuring SLE disease activity in previous 10 days, consisting 24 individual items in which signs and symptoms, laboratory tests, and physician's assessment for each item within each of 9 organ systems were given a weighted score (1 to 8 with higher score indicating increased activity) and summed if present at the time of the visit or in the preceding 10 days. The clinical SLEDAI-2K score was sum of 22 out of all 24 individual items from the SLEDAI-2K and ranges from 0 (no symptoms) to 101 (presence of all defined symptoms) with higher scores representing increased disease activity
Time Frame: Weeks 64, 80 and 104
Population: Modified Intent-to-Treat (MITT) Population
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Belimumab + Placebo | Belimumab + Rituximab | Belimumab + Standard Therapy
Number analyzed (Participants) | 72 | 144 | 47
Percentage of participants
  Week 64 | 5.6 [0.3 to 10.8] | 6.3 [2.3 to 10.2] | 10.6 [1.8 to 19.5]
  Week 80 | 4.2 [0 to 8.8] | 4.2 [0.9 to 7.4] | 12.8 [3.2 to 22.3]
  Week 104 | 1.4 [0 to 4.1] | 4.2 [0.9 to 7.4] | 6.4 [0 to 13.4]

6. Secondary Outcome: Percentage of Participants With a State of Complete Remission (CR) Sustained for at Least 24 Weeks During Week 52 to Week 104
Description: Percentage of participants with a state of CR (Principal Investigator [PI] assessed) was defined as percentage of participants with a SLEDAI-2K=0 achieved without immunosuppressants and with corticosteroids at prednisone equivalent dose of 0 mg/day,sustained for at least 24 weeks. Sustained CR was longest period a participant maintains CR without break calculated as last consecutive CR date minus first consecutive CR date plus 1. SLEDAI-2K consisted of 24 individual items within each 9 organ systems. Each item was given a weighted score (1 to 8, higher score indicates increased activity) and summed if present at time of visit or in preceding 10 days. SLEDAI-2K score was sum of all 24 individual items from SLEDAI-2K, ranges from 0(no symptoms) to 105(presence of all defined symptoms),higher scores indicates increased disease activity. Percentage of participants with a state of CR sustained for at least 24 weeks at any visit during Week 52 to Week 104 were reported.
Time Frame: Week 52 to Week 104
Population: Modified Intent-to-Treat (MITT) Population
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Belimumab + Placebo | Belimumab + Rituximab | Belimumab + Standard Therapy
Number analyzed (Participants) | 72 | 144 | 47
Percentage of participants | 2.8 [0 to 6.6] | 0 [NA to NA] — NA indicates that data was not available as confidence interval could not be calculated as there was no participant with a state of complete remission. | 6.4 [0 to 13.4]

7. Secondary Outcome: Percentage of Participants With a State of Clinical Remission (CLR) Sustained for at Least 24 Weeks From Week 80 to Week 104
Description: Percentage of participants with a state of CLR (PI assessed) at Week 104 was defined as percentage of participants with a clinical SLEDAI-2K score=0 (does not include anti-dsDNA and complement activity scores) achieved without immunosuppressants and with corticosteroids at a prednisone equivalent dose of 0 mg/day, sustained for at least 24 weeks(from Week 80 to Week 104). Sustained CLR is longest period a participant maintains CLR without a break, calculated as last consecutive CLR date minus first consecutive CLR date plus 1. SLEDAI-2K consisted of 24 individual items within each of 9 organ systems. Each item was given a weighted score(1 to 8 with higher score indicating increased activity) and summed if present at the time of visit or in preceding 10 days. The clinical SLEDAI-2K score was sum of 22 out of all 24 individual items from the SLEDAI-2K and ranges from 0 (no symptoms) to 101 (presence of all defined symptoms) with higher scores representing increased disease activity.
Time Frame: From Week 80 to Week 104
Population: Modified Intent-to-Treat (MITT) Population
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Belimumab + Placebo | Belimumab + Rituximab | Belimumab + Standard Therapy
Number analyzed (Participants) | 72 | 144 | 47
Percentage of participants | 2.8 [0 to 6.6] | 2.1 [0 to 4.4] | 4.3 [0 to 10.0]

8. Secondary Outcome: Percentage of Participants With a State of Complete Remission by Visits
Description: Percentage of participants with a state of complete remission (PI assessed) was defined as the percentage of participants with a SLEDAI-2K score =0, achieved without immunosuppressants and with corticosteroids at a prednisone equivalent dose of 0 mg/day. SLEDAI-2K was a weighted, cumulative index for measuring systemic lupus erythematosus (SLE) disease activity in the previous 10 days which consisted of 24 individual items in which signs and symptoms, laboratory tests, and physician's assessment for each item within for each of 9 organ systems were given a weighted score (1 to 8 with higher score indicating increased activity) and summed if present at the time of the visit or in the preceding 10 days. The SLEDAI-2K score was the sum of all 24 individual items from the SLEDAI-2K which ranges from 0 (no symptoms) to 105 (presence of all defined symptoms) with higher scores representing increased disease activity.
Time Frame: Weeks 60, 64, 72, 80, 88, 96 and 104
Population: Modified Intent-to-Treat (MITT) Population
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Belimumab + Placebo | Belimumab + Rituximab | Belimumab + Standard Therapy
Number analyzed (Participants) | 72 | 144 | 47
Percentage of participants
  Week 60 | 5.6 [0.3 to 10.8] | 0.7 [0 to 2.1] | 6.4 [0 to 13.4]
  Week 64 | 5.6 [0.3 to 10.8] | 0.7 [0 to 2.1] | 6.4 [0 to 13.4]
  Week 72 | 4.2 [0 to 8.8] | 0.7 [0 to 2.1] | 6.4 [0 to 13.4]
  Week 80 | 2.8 [0 to 6.6] | 1.4 [0 to 3.3] | 8.5 [0.5 to 16.5]
  Week 88 | 2.8 [0 to 6.6] | 0 [NA to NA] — NA indicates that data was not available as confidence interval could not be calculated as there was no participant with a state of complete remission. | 4.3 [0 to 10.0]
  Week 96 | 1.4 [0 to 4.1] | 0.7 [0 to 2.1] | 6.4 [0 to 13.4]
  Week 104 | 1.4 [0 to 4.1] | 0.7 [0 to 2.1] | 4.3 [0 to 10.0]

9. Secondary Outcome: Time to First Severe Flare
Description: Time to first severe SLE flare was the number of days from treatment start date until the participant met an event. Time to first severe flare was defined as event date minus treatment start date plus 1. Time to first severe flare was measured by Modified SLE flare index which identifies whether a participant had experienced a mild/moderate or severe flare. Analysis of first severe flare was performed on the modified SLE Flare index that excludes severe flares that were triggered only by an increase is SLEDAI-2K score to greater than 12.
Time Frame: Up to Week 104
Population: Modified Intent-to-Treat (MITT) Population
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Belimumab + Placebo | Belimumab + Rituximab | Belimumab + Standard Therapy
Number analyzed (Participants) | 72 | 144 | 47
Days | 372.0 [202.0 to 485.0] | 379.0 [198.0 to NA] — NA indicates that data was not available as only <75% of participants experienced the event within the treatment arm. Hence, third-quartile could not be derived. | 730.0 [210.0 to NA] — NA indicates that data was not available as only <75% of participants experienced the event within the treatment arm. Hence, third-quartile could not be derived.
Statistical Analysis 1: Comparison: Belimumab + Placebo vs Belimumab + Rituximab; Test type: Other; p = 0.2150, Cox proportional hazards model; Hazard Ratio (HR) = 0.81, 95% CI 2-sided [0.57 to 1.13] — Hazard ratio was calculated using Cox proportional hazards model with covariates: Baseline SLEDAI-2K, Baseline immunosuppressant, Baseline prednisone equivalent dose and treatment group. Belimumab + Standard therapy arm was excluded from model
Statistical Analysis 2: Comparison: Belimumab + Rituximab vs Belimumab + Standard Therapy; Test type: Other; Hazard Ratio (HR) = 1.64, 95% CI 2-sided [1.03 to 2.63] — Hazard ratio was calculated using Cox proportional hazards model with covariates: Baseline SLEDAI-2K, Baseline immunosuppressant, Baseline prednisone equivalent dose and treatment group. Belimumab + Placebo arm excluded from model

10. Secondary Outcome: Time to First Flare
Description: Time to first SLE flare was the number of days from treatment start date until the participant met an event. Time to first flare was defined as event date minus treatment start date plus 1. Time to first flare was measured by modified SLE flare index which identifies whether a participant had experienced a mild/moderate or severe flare.
Time Frame: Up to Week 104
Population: Modified Intent-to-Treat (MITT) Population
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Belimumab + Placebo | Belimumab + Rituximab | Belimumab + Standard Therapy
Number analyzed (Participants) | 72 | 144 | 47
Days | 168.0 [92.0 to 257.0] | 170.0 [57.0 to 365.0] | 168.0 [91.0 to 337.0]
Statistical Analysis 1: Comparison: Belimumab + Placebo vs Belimumab + Rituximab; Test type: Other; p = 0.3757, Cox proportional hazards model; Hazard Ratio (HR) = 0.87, 95% CI 2-sided [0.64 to 1.19] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 2: Comparison: Belimumab + Rituximab vs Belimumab + Standard Therapy; Test type: Other; Hazard Ratio (HR) = 1.03, 95% CI 2-sided [0.71 to 1.49] — [estimate comment as in outcome 9, analysis 2]

11. Secondary Outcome: Time to Disease Control Sustained for at Least 24 Weeks and Maintained Through Week 104
Description: Disease control sustained for at least 24 weeks and maintained through Week 104 was defined as SLEDAI-2K score <=2, achieved without immunosuppressants and with corticosteroids at a prednisone equivalent dose of <=5 mg/day. Time to disease control (PI assessed) was defined as the first visit of sustained disease control until Week 104 on or before Week 80 minus treatment start date (Day 1) plus 1. Sustained disease control was longest period a participant maintained disease control without a break. SLEDAI-2K consisted of 24 individual items within each of 9 organ systems. Each item was given a weighted score (1 to 8, higher score indicates increased activity) and summed if present at the time of visit or in preceding 10 days. SLEDAI-2K score was the sum of all 24 individual items from SLEDAI-2K , ranges from 0 (no symptoms) to 105 (presence of all defined symptoms),higher scores representing increased disease activity.
Time Frame: Up to Week 104
Population: Modified Intent-to-Treat (MITT) Population
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Belimumab + Placebo | Belimumab + Rituximab | Belimumab + Standard Therapy
Number analyzed (Participants) | 72 | 144 | 47
Days | NA [NA to NA] — NA indicates that data was not available as only <25% of participants experienced the event within the treatment arm. Hence, median and inter-quartile range could not be derived. | NA [NA to NA] — NA indicates that data was not available as only <25% of participants experienced the event within the treatment arm. Hence, median and inter-quartile range could not be derived. | NA [NA to NA] — NA indicates that data was not available as only <25% of participants experienced the event within the treatment arm. Hence, median and inter-quartile range could not be derived.
Statistical Analysis 1: Comparison: Belimumab + Placebo vs Belimumab + Rituximab; Test type: Other; p = 0.5127, Cox proportional hazards model; Hazard Ratio (HR) = 1.55, 95% CI 2-sided [0.42 to 5.78] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 2: Comparison: Belimumab + Rituximab vs Belimumab + Standard Therapy; Test type: Other; Hazard Ratio (HR) = 0.70, 95% CI 2-sided [0.23 to 2.10] — [estimate comment as in outcome 9, analysis 2]

12. Secondary Outcome: Time to Clinical Remission Sustained for at Least 24 Weeks and Maintained Through Week 104
Description: Clinical remission sustained for at least 24 weeks and maintained through Week 104 was defined as clinical SLEDAI-2K score=0 (does not include anti-dsDNA and complement activity scores), achieved without immunosuppressants and with corticosteroids at a prednisone equivalent dose of 0 mg/day. Time to CLR (PI assessed) was defined as first visit of sustained CLR until Week 104 on or before Week 80 minus treatment start date (Day 1) plus 1. Sustained CLR was longest period a participant maintained clinical remission without a break. SLEDAI-2K consisted of 24 individual items within each of 9 organ systems. Each item was given a weighted score (1 to 8, higher score indicates increased activity) and summed if present at the time of visit or in preceding 10 days. The clinical SLEDAI-2K score was sum of 22 out of all 24 individual items from the SLEDAI-2K and ranges from 0 (no symptoms) to 101 (presence of all defined symptoms) with higher scores representing increased disease activity.
Time Frame: Up to Week 104
Population: Modified Intent-to-Treat (MITT) Population
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Belimumab + Placebo | Belimumab + Rituximab | Belimumab + Standard Therapy
Number analyzed (Participants) | 72 | 144 | 47
Days | NA [NA to NA] — NA indicates that data was not available as only <25% of participants experienced the event within the treatment arm. Hence, median and inter-quartile range could not be derived. | NA [NA to NA] — NA indicates that data was not available as only <25% of participants experienced the event within the treatment arm. Hence, median and inter-quartile range could not be derived. | NA [NA to NA] — NA indicates that data was not available as only <25% of participants experienced the event within the treatment arm. Hence, median and inter-quartile range could not be derived.
Statistical Analysis 1: Comparison: Belimumab + Placebo vs Belimumab + Rituximab; Test type: Other; p = 0.8436, Cox proportional hazards model; Hazard Ratio (HR) = 0.83, 95% CI 2-sided [0.14 to 5.05] — Hazard ratio was calculated using Cox proportional hazards model with covariates: Baseline SLEDAI-2K, Baseline prednisone equivalent dose and treatment group. Belimumab + Standard therapy arm was excluded from model
Statistical Analysis 2: Comparison: Belimumab + Rituximab vs Belimumab + Standard Therapy; Test type: Other; Hazard Ratio (HR) = 0.52, 95% CI 2-sided [0.09 to 3.14] — Hazard ratio was calculated using Cox proportional hazards model with covariates: Baseline SLEDAI-2K, Baseline prednisone equivalent dose and treatment group. Belimumab + Placebo arm excluded from model

13. Secondary Outcome: Duration of Disease Control
Description: Duration of disease control was defined as SLEDAI-2K score <=2, achieved without immunosuppressants and with corticosteroids at a prednisone equivalent dose of <=5 mg/day. The duration of disease control (PI assessed) was the longest period between 2 visits that the participant was a disease control responder at all visits and calculated as the first visit of disease control minus last visit of disease control plus 1. SLEDAI-2K consisted of 24 individual items within each of 9 organ systems. Each item was given a weighted score (1 to 8, higher score indicates increased activity) and summed if present at the time of visit or in preceding 10 days. SLEDAI-2K score was the sum of all 24 individual items from SLEDAI-2K, ranges from 0(no symptoms) to 105 (presence of all defined symptoms),higher scores representing increased disease activity
Time Frame: Up to Week 104
Population: Modified Intent-to-Treat (MITT) Population. Only those participants with at least one assessment where disease control was met were analyzed.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Belimumab + Placebo | Belimumab + Rituximab | Belimumab + Standard Therapy
Number analyzed (Participants) | 34 | 77 | 31
Days | 49.5 [1.0 to 172.0] | 116.0 [21.0 to 265.0] | 116.0 [23.0 to 351.0]

14. Secondary Outcome: Duration of Clinical Remission
Description: Clinical remission was defined as clinical SLEDAI-2K score =0 (does not include anti-dsDNA and complement activity scores), achieved without immunosuppressants and with corticosteroids at a prednisone equivalent dose of 0 mg/day. The duration of clinical remission (PI assessed) was the longest period between 2 visits that the participant was a clinical remission responder at all visits and was calculated as the first visit of clinical remission minus last visit of clinical remission plus 1. SLEDAI-2K consisted of 24 individual items within each of 9 organ systems. Each item was given a weighted score (1 to 8, higher score indicates increased activity) and summed if present at the time of visit or in preceding 10 days. The clinical SLEDAI-2K score was sum of 22 out of all 24 individual items from the SLEDAI-2K and ranges from 0 (no symptoms) to 101 (presence of all defined symptoms) with higher scores representing increased disease activity.
Time Frame: Up to Week 104
Population: Modified Intent-to-Treat (MITT) Population. Only those participants with at least one assessment where clinical remission was met were analyzed.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Belimumab + Placebo | Belimumab + Rituximab | Belimumab + Standard Therapy
Number analyzed (Participants) | 13 | 22 | 11
Days | 31.0 [1.0 to 253.0] | 73.0 [29.0 to 225.0] | 176.0 [85.0 to 279.0]

15. Secondary Outcome: Change From Baseline in Systemic Lupus Erythematosus Disease Activity Index 2000 (SLEDAI-2K) Score by Visit (PI Assessed)
Description: The SLEDAI-2K consisted of 24 individual items within 9 organ systems. Each item was given a weighted score (1 to 8 with higher score indicating increased activity) and summed if present at the time of visit or in the preceding 10 days. Weighted scores for central nervous system (CNS) (7 items) was 8; for vascular (1 item) was 8; for Musculoskeletal (2 items) was 4; for Renal (4 items) was 4; for Mucocutaneous (3 items) was 2; for Cardiovascular and Respiratory (2 items) was 2; for Immunologic (2 items) was 2;for Constitutional (1 item) was 1 and for Hematologic (2 items) was 1. SLEDAI-2K score was the sum of all 24 individual items from the SLEDAI-2K which ranges from 0 (no symptoms) to 105 (presence of all defined symptoms) with higher scores representing increased disease activity. Baseline value was latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was defined as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1) and Weeks 4, 8, 12, 16, 20, 24, 26, 28, 32, 36, 40, 44, 48, 52, 60, 64, 72, 80, 88, 96, 104
Population: Modified Intent-to-Treat (MITT) Population. Only those participants with data available at specified time points were analyzed (represented by n=X in category titles).
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Belimumab + Placebo | Belimumab + Rituximab | Belimumab + Standard Therapy
Number analyzed (Participants) | 72 | 144 | 47
Scores on a scale
  Week 4; n=69, 137, 43: number analyzed (Participants) | 69 | 137 | 43
  Week 4; n=69, 137, 43 | -1.4 (2.75) | -0.8 (3.39) | -1.3 (3.15)
  Week 8; n=63, 132, 43: number analyzed (Participants) | 63 | 132 | 43
  Week 8; n=63, 132, 43 | -3.2 (3.59) | -2.9 (4.09) | -2.9 (3.43)
  Week 12; n=63, 131, 43: number analyzed (Participants) | 63 | 131 | 43
  Week 12; n=63, 131, 43 | -2.8 (3.50) | -3.6 (4.32) | -2.9 (3.68)
  Week 16; n=65, 129, 43: number analyzed (Participants) | 65 | 129 | 43
  Week 16; n=65, 129, 43 | -3.4 (4.12) | -4.4 (4.62) | -4.1 (3.29)
  Week 20; n=63, 127, 44: number analyzed (Participants) | 63 | 127 | 44
  Week 20; n=63, 127, 44 | -3.8 (4.06) | -5.0 (4.44) | -3.8 (3.98)
  Week 24; n=61, 128, 43: number analyzed (Participants) | 61 | 128 | 43
  Week 24; n=61, 128, 43 | -4.0 (3.71) | -5.0 (4.45) | -5.0 (4.00)
  Week 26; n=61, 118, 40: number analyzed (Participants) | 61 | 118 | 40
  Week 26; n=61, 118, 40 | -4.1 (3.61) | -5.4 (4.79) | -5.0 (3.18)
  Week 28; n=62, 125, 43: number analyzed (Participants) | 62 | 125 | 43
  Week 28; n=62, 125, 43 | -3.7 (3.79) | -5.1 (4.74) | -5.2 (4.31)
  Week 32; n=61, 125, 43: number analyzed (Participants) | 61 | 125 | 43
  Week 32; n=61, 125, 43 | -4.7 (3.87) | -5.7 (5.03) | -5.3 (3.90)
  Week 36; n=61, 125, 43: number analyzed (Participants) | 61 | 125 | 43
  Week 36; n=61, 125, 43 | -5.0 (4.43) | -5.6 (5.21) | -5.0 (3.68)
  Week 40; n=62, 125, 43: number analyzed (Participants) | 62 | 125 | 43
  Week 40; n=62, 125, 43 | -4.6 (4.14) | -5.8 (4.83) | -5.0 (3.78)
  Week 44; n=62, 122, 43: number analyzed (Participants) | 62 | 122 | 43
  Week 44; n=62, 122, 43 | -4.7 (4.71) | -6.1 (4.47) | -5.2 (4.06)
  Week 48; n=59, 122, 40: number analyzed (Participants) | 59 | 122 | 40
  Week 48; n=59, 122, 40 | -4.5 (4.16) | -6.2 (4.59) | -5.3 (4.08)
  Week 52; n=62, 119, 39: number analyzed (Participants) | 62 | 119 | 39
  Week 52; n=62, 119, 39 | -5.3 (4.62) | -6.1 (4.42) | -5.6 (4.02)
  Week 60; n=57, 114, 37: number analyzed (Participants) | 57 | 114 | 37
  Week 60; n=57, 114, 37 | -5.0 (4.15) | -5.8 (5.17) | -6.0 (3.94)
  Week 64; n=60, 117, 36: number analyzed (Participants) | 60 | 117 | 36
  Week 64; n=60, 117, 36 | -5.1 (4.16) | -6.2 (4.96) | -5.5 (4.40)
  Week 72; n=49, 103, 30: number analyzed (Participants) | 49 | 103 | 30
  Week 72; n=49, 103, 30 | -5.2 (4.32) | -6.6 (4.50) | -5.3 (4.63)
  Week 80; n=46, 102, 36: number analyzed (Participants) | 46 | 102 | 36
  Week 80; n=46, 102, 36 | -5.4 (4.58) | -6.5 (4.79) | -6.0 (4.08)
  Week 88; n=49, 101, 34: number analyzed (Participants) | 49 | 101 | 34
  Week 88; n=49, 101, 34 | -5.3 (4.61) | -6.5 (4.29) | -6.1 (3.80)
  Week 96; n=49, 100, 34: number analyzed (Participants) | 49 | 100 | 34
  Week 96; n=49, 100, 34 | -5.6 (4.35) | -7.0 (4.44) | -6.1 (3.80)
  Week 104; n=50, 104, 34: number analyzed (Participants) | 50 | 104 | 34
  Week 104; n=50, 104, 34 | -5.1 (3.69) | -7.2 (4.22) | -6.3 (3.76)

16. Secondary Outcome: Percentage of Participants With SLEDAI-2K Organ Improvement Compared to Baseline by Visits (PI Assessed)
Description: SLEDAI-2K assessments consisted of 24 individual items with 9 organ systems. Each item was given a weighted score(1 to 8 with higher score indicating increased activity)and summed if present at the time of analysis. SLEDAI-2K score was sum of all 24 individual items from SLEDAI-2K ranges from 0(no symptoms) to 105(presence of all defined symptoms). Higher scores indicates increased disease activity. An improvement was defined as a decrease(compared to Baseline) in SLEDAI-2K score within same organ system at a post-Baseline visit. Baseline value was latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Data for following organ systems was reported: CNS total, Vascular total, Musculoskeletal total, Renal total, Mucocutaneous total, Cardiovascular (Cardio) and Respiratory (Resp) total, Immunologic total and Hematologic total. Constitutional organ system was removed from analysis and its one item (fever)moved to hematologic organ system.
Time Frame: Baseline (Day 1) and Weeks 4, 8, 12, 16, 20, 24, 26, 28, 32, 36, 40, 44, 48, 52, 60, 64, 72, 80, 88, 96, 104
Population: Modified Intent-to-Treat (MITT) Population. Only those participants with data available at specified time points were analyzed (represented by n=X in category titles). Only participants with organ system involvement at Baseline were included.
Measure: Number; unit: Percentage of participants
Arm/Group | Belimumab + Placebo | Belimumab + Rituximab | Belimumab + Standard Therapy
Number analyzed (Participants) | 72 | 144 | 47
Percentage of participants
  CNS Total; Week 4; n= 2,3,2: number analyzed (Participants) | 2 | 3 | 2
  CNS Total; Week 4; n= 2,3,2 | 0 | 33.3 | 0
  CNS Total; Week 8; n= 2,3,2: number analyzed (Participants) | 2 | 3 | 2
  CNS Total; Week 8; n= 2,3,2 | 50.0 | 66.7 | 0
  CNS Total; Week 12; n= 2,3,2: number analyzed (Participants) | 2 | 3 | 2
  CNS Total; Week 12; n= 2,3,2 | 50.0 | 66.7 | 50.0
  CNS Total; Week 16; n= 2,3,2: number analyzed (Participants) | 2 | 3 | 2
  CNS Total; Week 16; n= 2,3,2 | 50.0 | 66.7 | 0
  CNS Total; Week 20; n= 2,3,2: number analyzed (Participants) | 2 | 3 | 2
  CNS Total; Week 20; n= 2,3,2 | 100 | 66.7 | 0
  CNS Total; Week 24; n= 2,3,2: number analyzed (Participants) | 2 | 3 | 2
  CNS Total; Week 24; n= 2,3,2 | 100 | 66.7 | 100
  CNS Total; Week 26; n= 2,3,2: number analyzed (Participants) | 2 | 3 | 2
  CNS Total; Week 26; n= 2,3,2 | 50.0 | 66.7 | 0
  CNS Total; Week 28; n= 2,3,2: number analyzed (Participants) | 2 | 3 | 2
  CNS Total; Week 28; n= 2,3,2 | 100 | 66.7 | 100
  CNS Total; Week 32; n= 2,3,2: number analyzed (Participants) | 2 | 3 | 2
  CNS Total; Week 32; n= 2,3,2 | 100 | 66.7 | 100
  CNS Total; Week 36; n= 2,3,2: number analyzed (Participants) | 2 | 3 | 2
  CNS Total; Week 36; n= 2,3,2 | 100 | 66.7 | 50.0
  CNS Total; Week 40; n= 2,3,2: number analyzed (Participants) | 2 | 3 | 2
  CNS Total; Week 40; n= 2,3,2 | 100 | 66.7 | 100
  CNS Total; Week 44; n= 2,3,2: number analyzed (Participants) | 2 | 3 | 2
  CNS Total; Week 44; n= 2,3,2 | 100 | 66.7 | 100
  CNS Total; Week 48; n= 2,3,2: number analyzed (Participants) | 2 | 3 | 2
  CNS Total; Week 48; n= 2,3,2 | 100 | 66.7 | 50.0
  CNS Total; Week 52; n= 2,3,2: number analyzed (Participants) | 2 | 3 | 2
  CNS Total; Week 52; n= 2,3,2 | 100 | 66.7 | 100
  CNS Total; Week 60; n= 2,3,2: number analyzed (Participants) | 2 | 3 | 2
  CNS Total; Week 60; n= 2,3,2 | 100 | 66.7 | 100
  CNS Total; Week 64; n= 2,3,2: number analyzed (Participants) | 2 | 3 | 2
  CNS Total; Week 64; n= 2,3,2 | 100 | 66.7 | 100
  CNS Total; Week 72; n= 2,3,2: number analyzed (Participants) | 2 | 3 | 2
  CNS Total; Week 72; n= 2,3,2 | 100 | 33.3 | 50.0
  CNS Total; Week 80; n= 2,3,2: number analyzed (Participants) | 2 | 3 | 2
  CNS Total; Week 80; n= 2,3,2 | 100 | 33.3 | 50.0
  CNS Total; Week 88; n= 2,3,2: number analyzed (Participants) | 2 | 3 | 2
  CNS Total; Week 88; n= 2,3,2 | 100 | 33.3 | 100
  CNS Total; Week 96; n= 2,3,2: number analyzed (Participants) | 2 | 3 | 2
  CNS Total; Week 96; n= 2,3,2 | 100 | 33.3 | 100
  CNS Total; Week 104; n=2,3,2: number analyzed (Participants) | 2 | 3 | 2
  CNS Total; Week 104; n=2,3,2 | 100 | 33.3 | 100
  Vascular Total; Week 4; n= 6,11,0: number analyzed (Participants) | 6 | 11 | 0
  Vascular Total; Week 4; n= 6,11,0 | 50.0 | 9.1 |
  Vascular Total; Week 8; n= 6,11,0: number analyzed (Participants) | 6 | 11 | 0
  Vascular Total; Week 8; n= 6,11,0 | 33.3 | 36.4 |
  Vascular Total; Week 12; n= 6,11,0: number analyzed (Participants) | 6 | 11 | 0
  Vascular Total; Week 12; n= 6,11,0 | 50.0 | 54.5 |
  Vascular Total; Week 16; n= 6,11,0: number analyzed (Participants) | 6 | 11 | 0
  Vascular Total; Week 16; n= 6,11,0 | 50.0 | 54.5 |
  Vascular Total; Week 20; n=6,11,0: number analyzed (Participants) | 6 | 11 | 0
  Vascular Total; Week 20; n=6,11,0 | 50.0 | 72.7 |
  Vascular Total; Week 24; n= 6,11,0: number analyzed (Participants) | 6 | 11 | 0
  Vascular Total; Week 24; n= 6,11,0 | 50.0 | 72.7 |
  Vascular Total; Week 26; n= 6, 11, 0: number analyzed (Participants) | 6 | 11 | 0
  Vascular Total; Week 26; n= 6, 11, 0 | 50.0 | 63.6 |
  Vascular Total; Week 28; n= 6, 11,0: number analyzed (Participants) | 6 | 11 | 0
  Vascular Total; Week 28; n= 6, 11,0 | 33.3 | 72.7 |
  Vascular Total; Week 32; n= 6,11, 0: number analyzed (Participants) | 6 | 11 | 0
  Vascular Total; Week 32; n= 6,11, 0 | 50.0 | 72.7 |
  Vascular Total; Week 36; n= 6, 11,0: number analyzed (Participants) | 6 | 11 | 0
  Vascular Total; Week 36; n= 6, 11,0 | 50.0 | 63.6 |
  Vascular Total; Week 40; n= 6, 11,0: number analyzed (Participants) | 6 | 11 | 0
  Vascular Total; Week 40; n= 6, 11,0 | 33.3 | 72.7 |
  Vascular Total; Week 44; n= 6, 11, 0: number analyzed (Participants) | 6 | 11 | 0
  Vascular Total; Week 44; n= 6, 11, 0 | 33.3 | 72.7 |
  Vascular Total; Week 48; n= 6, 11, 0: number analyzed (Participants) | 6 | 11 | 0
  Vascular Total; Week 48; n= 6, 11, 0 | 33.3 | 63.6 |
  Vascular Total; Week 52; n= 6, 11, 0: number analyzed (Participants) | 6 | 11 | 0
  Vascular Total; Week 52; n= 6, 11, 0 | 66.7 | 63.6 |
  Vascular Total; Week 60; n= 6, 11, 0: number analyzed (Participants) | 6 | 11 | 0
  Vascular Total; Week 60; n= 6, 11, 0 | 50.0 | 63.6 |
  Vascular Total; Week 64; n= 6, 11, 0: number analyzed (Participants) | 6 | 11 | 0
  Vascular Total; Week 64; n= 6, 11, 0 | 50.0 | 90.9 |
  Vascular Total; Week 72; n= 6, 11, 0: number analyzed (Participants) | 6 | 11 | 0
  Vascular Total; Week 72; n= 6, 11, 0 | 33.3 | 81.8 |
  Vascular Total; Week 80; n= 6, 11, 0: number analyzed (Participants) | 6 | 11 | 0
  Vascular Total; Week 80; n= 6, 11, 0 | 50.0 | 72.7 |
  Vascular Total; Week 88; n= 6, 11, 0: number analyzed (Participants) | 6 | 11 | 0
  Vascular Total; Week 88; n= 6, 11, 0 | 50.0 | 45.5 |
  Vascular Total; Week 96; n= 6, 11, 0: number analyzed (Participants) | 6 | 11 | 0
  Vascular Total; Week 96; n= 6, 11, 0 | 50.0 | 63.6 |
  Vascular Total; Week 104; n= 6, 11, 0: number analyzed (Participants) | 6 | 11 | 0
  Vascular Total; Week 104; n= 6, 11, 0 | 33.3 | 72.7 |
  Musculoskeletal Total; Week 4; n= 57, 110, 34: number analyzed (Participants) | 57 | 110 | 34
  Musculoskeletal Total; Week 4; n= 57, 110, 34 | 22.8 | 13.6 | 23.5
  Musculoskeletal Total; Week 8; n=57,110, 34: number analyzed (Participants) | 57 | 110 | 34
  Musculoskeletal Total; Week 8; n=57,110, 34 | 40.4 | 40.0 | 50.0
  Musculoskeletal Total; Week 12; n= 57,110,34: number analyzed (Participants) | 57 | 110 | 34
  Musculoskeletal Total; Week 12; n= 57,110,34 | 36.8 | 44.5 | 47.1
  Musculoskeletal Total; Week 16; n= 57,110,34: number analyzed (Participants) | 57 | 110 | 34
  Musculoskeletal Total; Week 16; n= 57,110,34 | 42.1 | 56.4 | 67.6
  Musculoskeletal Total; Week 20; n= 57,110,34: number analyzed (Participants) | 57 | 110 | 34
  Musculoskeletal Total; Week 20; n= 57,110,34 | 47.4 | 58.2 | 64.7
  Musculoskeletal Total; Week 24; n= 57,110,34: number analyzed (Participants) | 57 | 110 | 34
  Musculoskeletal Total; Week 24; n= 57,110,34 | 42.1 | 54.5 | 70.6
  Musculoskeletal Total;; Week 26; n=57,110,34: number analyzed (Participants) | 57 | 110 | 34
  Musculoskeletal Total;; Week 26; n=57,110,34 | 43.9 | 46.4 | 73.5
  Musculoskeletal Total; Week 28; n= 57,110,34: number analyzed (Participants) | 57 | 110 | 34
  Musculoskeletal Total; Week 28; n= 57,110,34 | 49.1 | 53.6 | 76.5
  Musculoskeletal Total; Week 32; n= 57,110,34: number analyzed (Participants) | 57 | 110 | 34
  Musculoskeletal Total; Week 32; n= 57,110,34 | 54.4 | 63.6 | 76.5
  Musculoskeletal Total; Week 36; n= 57,110,34: number analyzed (Participants) | 57 | 110 | 34
  Musculoskeletal Total; Week 36; n= 57,110,34 | 61.4 | 61.8 | 76.5
  Musculoskeletal Total; Week 40; n= 57,110,34: number analyzed (Participants) | 57 | 110 | 34
  Musculoskeletal Total; Week 40; n= 57,110,34 | 54.4 | 58.2 | 73.5
  Musculoskeletal Total; Week 44; n= 57,110,34: number analyzed (Participants) | 57 | 110 | 34
  Musculoskeletal Total; Week 44; n= 57,110,34 | 50.9 | 60.0 | 76.5
  Musculoskeletal Total; Week 48; n= 57,110,34: number analyzed (Participants) | 57 | 110 | 34
  Musculoskeletal Total; Week 48; n= 57,110,34 | 57.9 | 60.9 | 73.5
  Musculoskeletal Total; Week 52; n= 57,110,34: number analyzed (Participants) | 57 | 110 | 34
  Musculoskeletal Total; Week 52; n= 57,110,34 | 59.6 | 59.1 | 73.5
  Musculoskeletal Total; Week 60; n= 57,110,34: number analyzed (Participants) | 57 | 110 | 34
  Musculoskeletal Total; Week 60; n= 57,110,34 | 54.4 | 54.5 | 67.6
  Musculoskeletal Total; Week 64; n= 57,110,34: number analyzed (Participants) | 57 | 110 | 34
  Musculoskeletal Total; Week 64; n= 57,110,34 | 56.1 | 55.5 | 67.6
  Musculoskeletal Total; Week 72; n= 57,110,34: number analyzed (Participants) | 57 | 110 | 34
  Musculoskeletal Total; Week 72; n= 57,110,34 | 47.4 | 58.2 | 58.8
  Musculoskeletal Total; Week 80; n= 57,110,34: number analyzed (Participants) | 57 | 110 | 34
  Musculoskeletal Total; Week 80; n= 57,110,34 | 47.4 | 58.2 | 76.5
  Musculoskeletal Total; Week 88; n= 57,110,34: number analyzed (Participants) | 57 | 110 | 34
  Musculoskeletal Total; Week 88; n= 57,110,34 | 57.9 | 59.1 | 67.6
  Musculoskeletal Total; Week 96; n= 57,110,34: number analyzed (Participants) | 57 | 110 | 34
  Musculoskeletal Total; Week 96; n= 57,110,34 | 50.9 | 60.9 | 70.6
  Musculoskeletal Total; Week 104; n= 57,110,34: number analyzed (Participants) | 57 | 110 | 34
  Musculoskeletal Total; Week 104; n= 57,110,34 | 47.4 | 64.5 | 67.6
  Renal Total; Week 4; n= 14,23,8: number analyzed (Participants) | 14 | 23 | 8
  Renal Total; Week 4; n= 14,23,8 | 21.4 | 30.4 | 12.5
  Renal Total; Week 8; n= 14, 23, 8: number analyzed (Participants) | 14 | 23 | 8
  Renal Total; Week 8; n= 14, 23, 8 | 50.0 | 43.5 | 12.5
  Renal Total; Week 12; n= 14, 23, 8: number analyzed (Participants) | 14 | 23 | 8
  Renal Total; Week 12; n= 14, 23, 8 | 28.6 | 52.2 | 12.5
  Renal Total; Week 16; n= 14, 23, 8: number analyzed (Participants) | 14 | 23 | 8
  Renal Total; Week 16; n= 14, 23, 8 | 35.7 | 52.2 | 12.5
  Renal Total; Week 20; n= 14, 23, 8: number analyzed (Participants) | 14 | 23 | 8
  Renal Total; Week 20; n= 14, 23, 8 | 57.1 | 60.9 | 12.5
  Renal Total; Week 24; n= 14, 23, 8: number analyzed (Participants) | 14 | 23 | 8
  Renal Total; Week 24; n= 14, 23, 8 | 35.7 | 60.9 | 12.5
  Renal Total; Week 26; n= 14, 23, 8: number analyzed (Participants) | 14 | 23 | 8
  Renal Total; Week 26; n= 14, 23, 8 | 28.6 | 65.2 | 25.0
  Renal Total; Week 28; n= 14, 23, 8: number analyzed (Participants) | 14 | 23 | 8
  Renal Total; Week 28; n= 14, 23, 8 | 21.4 | 56.5 | 37.5
  Renal Total; Week 32; n= 14, 23, 8: number analyzed (Participants) | 14 | 23 | 8
  Renal Total; Week 32; n= 14, 23, 8 | 35.7 | 65.2 | 25.0
  Renal Total; Week 36; n= 14, 23, 8: number analyzed (Participants) | 14 | 23 | 8
  Renal Total; Week 36; n= 14, 23, 8 | 42.9 | 65.2 | 50.0
  Renal Total; Week 40; n=14, 23, 8: number analyzed (Participants) | 14 | 23 | 8
  Renal Total; Week 40; n=14, 23, 8 | 42.9 | 69.6 | 25.0
  Renal Total; Week 44; n= 14, 23, 8: number analyzed (Participants) | 14 | 23 | 8
  Renal Total; Week 44; n= 14, 23, 8 | 50.0 | 69.6 | 12.5
  Renal Total; Week 48; n=14, 23, 8: number analyzed (Participants) | 14 | 23 | 8
  Renal Total; Week 48; n=14, 23, 8 | 42.9 | 69.6 | 50.0
  Renal Total; Week 52; n= 14, 23, 8: number analyzed (Participants) | 14 | 23 | 8
  Renal Total; Week 52; n= 14, 23, 8 | 64.3 | 69.6 | 25.0
  Renal Total; Week 60; n= 14, 23, 8: number analyzed (Participants) | 14 | 23 | 8
  Renal Total; Week 60; n= 14, 23, 8 | 50.0 | 65.2 | 25.0
  Renal Total; Week 64; n= 14, 23, 8: number analyzed (Participants) | 14 | 23 | 8
  Renal Total; Week 64; n= 14, 23, 8 | 50.0 | 69.6 | 12.5
  Renal Total; Week 72; n= 14, 23, 8: number analyzed (Participants) | 14 | 23 | 8
  Renal Total; Week 72; n= 14, 23, 8 | 50.0 | 65.2 | 12.5
  Renal Total; Week 80; n= 14, 23, 8: number analyzed (Participants) | 14 | 23 | 8
  Renal Total; Week 80; n= 14, 23, 8 | 42.9 | 65.2 | 50.0
  Renal Total; Week 88; n= 14, 23, 8: number analyzed (Participants) | 14 | 23 | 8
  Renal Total; Week 88; n= 14, 23, 8 | 50.0 | 73.9 | 25.0
  Renal Total; Week 96; n= 14, 23, 8: number analyzed (Participants) | 14 | 23 | 8
  Renal Total; Week 96; n= 14, 23, 8 | 35.7 | 78.3 | 37.5
  Renal Total; Week 104; n= 14, 23, 8: number analyzed (Participants) | 14 | 23 | 8
  Renal Total; Week 104; n= 14, 23, 8 | 35.7 | 69.6 | 50.0
  Mucocutaneous Total; Week 4; n= 59, 126,43: number analyzed (Participants) | 59 | 126 | 43
  Mucocutaneous Total; Week 4; n= 59, 126,43 | 30.5 | 28.6 | 32.6
  Mucocutaneous Total; Week 8; n= 59,126,43: number analyzed (Participants) | 59 | 126 | 43
  Mucocutaneous Total; Week 8; n= 59,126,43 | 54.2 | 45.2 | 51.2
  Mucocutaneous Total; Week 12; n= 59, 126, 43: number analyzed (Participants) | 59 | 126 | 43
  Mucocutaneous Total; Week 12; n= 59, 126, 43 | 55.9 | 57.1 | 55.8
  Mucocutaneous Total; Week 16; n= 59, 126, 43: number analyzed (Participants) | 59 | 126 | 43
  Mucocutaneous Total; Week 16; n= 59, 126, 43 | 57.6 | 58.7 | 67.4
  Mucocutaneous Total; Week 20; n= 59, 126, 43: number analyzed (Participants) | 59 | 126 | 43
  Mucocutaneous Total; Week 20; n= 59, 126, 43 | 50.8 | 62.7 | 69.8
  Mucocutaneous Total; Week 24; n= 59, 126, 43: number analyzed (Participants) | 59 | 126 | 43
  Mucocutaneous Total; Week 24; n= 59, 126, 43 | 59.3 | 61.9 | 69.8
  Mucocutaneous Total; Week 26; n=59, 126, 43: number analyzed (Participants) | 59 | 126 | 43
  Mucocutaneous Total; Week 26; n=59, 126, 43 | 59.3 | 60.3 | 65.1
  Mucocutaneous Total; Week 28; n= 59, 126, 43: number analyzed (Participants) | 59 | 126 | 43
  Mucocutaneous Total; Week 28; n= 59, 126, 43 | 62.7 | 62.7 | 69.8
  Mucocutaneous Total; Week 32; n= 59, 126, 43: number analyzed (Participants) | 59 | 126 | 43
  Mucocutaneous Total; Week 32; n= 59, 126, 43 | 62.7 | 65.1 | 74.4
  Mucocutaneous Total; Week 36; n= 59, 126, 43: number analyzed (Participants) | 59 | 126 | 43
  Mucocutaneous Total; Week 36; n= 59, 126, 43 | 66.1 | 65.9 | 69.8
  Mucocutaneous Total; Week 40; n= 59, 126, 43: number analyzed (Participants) | 59 | 126 | 43
  Mucocutaneous Total; Week 40; n= 59, 126, 43 | 62.7 | 66.7 | 67.4
  Mucocutaneous Total; Week 44; n= 59, 126, 43: number analyzed (Participants) | 59 | 126 | 43
  Mucocutaneous Total; Week 44; n= 59, 126, 43 | 61.0 | 61.1 | 69.8
  Mucocutaneous Total; Week 48; n= 59, 126, 43: number analyzed (Participants) | 59 | 126 | 43
  Mucocutaneous Total; Week 48; n= 59, 126, 43 | 50.8 | 66.7 | 69.8
  Mucocutaneous Total; Week 52; n=59, 126, 43: number analyzed (Participants) | 59 | 126 | 43
  Mucocutaneous Total; Week 52; n=59, 126, 43 | 64.4 | 64.3 | 69.8
  Mucocutaneous Total; Week 60; n=59, 126, 43: number analyzed (Participants) | 59 | 126 | 43
  Mucocutaneous Total; Week 60; n=59, 126, 43 | 55.9 | 65.1 | 67.4
  Mucocutaneous Total; Week 64; n=59, 126, 43: number analyzed (Participants) | 59 | 126 | 43
  Mucocutaneous Total; Week 64; n=59, 126, 43 | 64.4 | 65.9 | 62.8
  Mucocutaneous Total; Week 72; n=59, 126, 43: number analyzed (Participants) | 59 | 126 | 43
  Mucocutaneous Total; Week 72; n=59, 126, 43 | 57.6 | 60.3 | 58.1
  Mucocutaneous Total; Week 80; n= 59, 126, 43: number analyzed (Participants) | 59 | 126 | 43
  Mucocutaneous Total; Week 80; n= 59, 126, 43 | 62.7 | 61.9 | 62.8
  Mucocutaneous Total; Week 88; n= 59, 126, 43: number analyzed (Participants) | 59 | 126 | 43
  Mucocutaneous Total; Week 88; n= 59, 126, 43 | 59.3 | 62.7 | 67.4
  Mucocutaneous Total; Week 96; n= 59, 126, 43: number analyzed (Participants) | 59 | 126 | 43
  Mucocutaneous Total; Week 96; n= 59, 126, 43 | 52.5 | 62.7 | 62.7
  Mucocutaneous Total; Week 104; n= 59, 126, 43: number analyzed (Participants) | 59 | 126 | 43
  Mucocutaneous Total; Week 104; n= 59, 126, 43 | 61.0 | 69.0 | 60.5
  Cardio and Resp Total; Week 4; n= 3, 7, 0: number analyzed (Participants) | 3 | 7 | 0
  Cardio and Resp Total; Week 4; n= 3, 7, 0 | 0 | 42.9 |
  Cardio and Resp Total; Week 8; n= 3, 7, 0: number analyzed (Participants) | 3 | 7 | 0
  Cardio and Resp Total; Week 8; n= 3, 7, 0 | 0 | 71.4 |
  Cardio and Resp Total; Week 12; n= 3, 7, 0: number analyzed (Participants) | 3 | 7 | 0
  Cardio and Resp Total; Week 12; n= 3, 7, 0 | 0 | 71.4 |
  Cardio and Resp Total; Week 16; n= 3, 7, 0: number analyzed (Participants) | 3 | 7 | 0
  Cardio and Resp Total; Week 16; n= 3, 7, 0 | 0 | 85.7 |
  Cardio and Resp Total; Week 20; n= 3,7, 0: number analyzed (Participants) | 3 | 7 | 0
  Cardio and Resp Total; Week 20; n= 3,7, 0 | 33.3 | 71.4 |
  Cardio and Resp Total; Week 24; n= 3, 7, 0: number analyzed (Participants) | 3 | 7 | 0
  Cardio and Resp Total; Week 24; n= 3, 7, 0 | 66.7 | 100 |
  Cardio and Resp Total; Week 26; n=3, 7, 0: number analyzed (Participants) | 3 | 7 | 0
  Cardio and Resp Total; Week 26; n=3, 7, 0 | 0 | 85.7 |
  Cardio and Resp Total; Week 28; n= 3,7, 0: number analyzed (Participants) | 3 | 7 | 0
  Cardio and Resp Total; Week 28; n= 3,7, 0 | 0 | 85.7 |
  Cardio and Resp Total; Week 32; n= 3, 7, 0: number analyzed (Participants) | 3 | 7 | 0
  Cardio and Resp Total; Week 32; n= 3, 7, 0 | 33.3 | 100 |
  Cardio and Resp Total; Week 36; n= 3, 7, 0: number analyzed (Participants) | 3 | 7 | 0
  Cardio and Resp Total; Week 36; n= 3, 7, 0 | 66.7 | 85.7 |
  Cardio and Resp Total; Week 40; n=3,7, 0: number analyzed (Participants) | 3 | 7 | 0
  Cardio and Resp Total; Week 40; n=3,7, 0 | 33.3 | 71.4 |
  Cardio and Resp Total; Week 44; n= 3,7, 0: number analyzed (Participants) | 3 | 7 | 0
  Cardio and Resp Total; Week 44; n= 3,7, 0 | 66.7 | 57.1 |
  Cardio and Resp Total; Week 48; n= 3, 7, 0: number analyzed (Participants) | 3 | 7 | 0
  Cardio and Resp Total; Week 48; n= 3, 7, 0 | 33.3 | 85.7 |
  Cardio and Resp Total; Week 52; n= 3, 7, 0: number analyzed (Participants) | 3 | 7 | 0
  Cardio and Resp Total; Week 52; n= 3, 7, 0 | 66.7 | 85.7 |
  Cardio and Resp Total; Week 60; n= 3,7,0: number analyzed (Participants) | 3 | 7 | 0
  Cardio and Resp Total; Week 60; n= 3,7,0 | 100 | 71.4 |
  Cardio and Resp Total; Week 64; n=3,7,0: number analyzed (Participants) | 3 | 7 | 0
  Cardio and Resp Total; Week 64; n=3,7,0 | 100 | 85.7 |
  Cardio and Resp Total; Week 72; n= 3,7,0: number analyzed (Participants) | 3 | 7 | 0
  Cardio and Resp Total; Week 72; n= 3,7,0 | 66.7 | 71.4 |
  Cardio and Resp Total; Week 80; n=3,7,0: number analyzed (Participants) | 3 | 7 | 0
  Cardio and Resp Total; Week 80; n=3,7,0 | 66.7 | 85.7 |
  Cardio and Resp Total; Week 88; n= 3,7,0: number analyzed (Participants) | 3 | 7 | 0
  Cardio and Resp Total; Week 88; n= 3,7,0 | 66.7 | 71.4 |
  Cardio and Resp Total; Week 96; n= 3,7,0: number analyzed (Participants) | 3 | 7 | 0
  Cardio and Resp Total; Week 96; n= 3,7,0 | 66.7 | 71.4 |
  Cardio and Resp Total; Week 104; n= 3,7,0: number analyzed (Participants) | 3 | 7 | 0
  Cardio and Resp Total; Week 104; n= 3,7,0 | 66.7 | 71.4 |
  Immunologic Total; Week 4; n=48, 104, 34: number analyzed (Participants) | 48 | 104 | 34
  Immunologic Total; Week 4; n=48, 104, 34 | 12.5 | 10.6 | 17.6
  Immunologic Total; Week 8; n= 48, 104, 34: number analyzed (Participants) | 48 | 104 | 34
  Immunologic Total; Week 8; n= 48, 104, 34 | 16.7 | 17.3 | 17.6
  Immunologic Total; Week 12; n= 48, 104, 34: number analyzed (Participants) | 48 | 104 | 34
  Immunologic Total; Week 12; n= 48, 104, 34 | 22.9 | 24.0 | 17.6
  Immunologic Total; Week 16; n= 48, 104, 34: number analyzed (Participants) | 48 | 104 | 34
  Immunologic Total; Week 16; n= 48, 104, 34 | 20.8 | 30.8 | 11.8
  Immunologic Total; Week 20; n= 48, 104, 34: number analyzed (Participants) | 48 | 104 | 34
  Immunologic Total; Week 20; n= 48, 104, 34 | 20.8 | 36.5 | 23.5
  Immunologic Total; Week 24; n= 48, 104, 34: number analyzed (Participants) | 48 | 104 | 34
  Immunologic Total; Week 24; n= 48, 104, 34 | 22.9 | 34.6 | 20.6
  Immunologic Total; Week 26; n= 48, 104, 34: number analyzed (Participants) | 48 | 104 | 34
  Immunologic Total; Week 26; n= 48, 104, 34 | 18.8 | 39.4 | 11.8
  Immunologic Total; Week 28; n= 48, 104, 34: number analyzed (Participants) | 48 | 104 | 34
  Immunologic Total; Week 28; n= 48, 104, 34 | 18.8 | 34.6 | 20.6
  Immunologic Total; Week 32; n= 48, 104, 34: number analyzed (Participants) | 48 | 104 | 34
  Immunologic Total; Week 32; n= 48, 104, 34 | 25.0 | 40.4 | 23.5
  Immunologic Total; Week 36; n= 48, 104, 34: number analyzed (Participants) | 48 | 104 | 34
  Immunologic Total; Week 36; n= 48, 104, 34 | 20.8 | 41.3 | 17.6
  Immunologic Total; Week 40; n= 48, 104, 34: number analyzed (Participants) | 48 | 104 | 34
  Immunologic Total; Week 40; n= 48, 104, 34 | 14.6 | 44.2 | 23.5
  Immunologic Total; Week 44; n= 48, 104, 34: number analyzed (Participants) | 48 | 104 | 34
  Immunologic Total; Week 44; n= 48, 104, 34 | 25.0 | 39.4 | 38.2
  Immunologic Total; Week 48; n= 48, 104, 34: number analyzed (Participants) | 48 | 104 | 34
  Immunologic Total; Week 48; n= 48, 104, 34 | 20.8 | 41.3 | 29.4
  Immunologic Total; Week 52; n= 48, 104, 34: number analyzed (Participants) | 48 | 104 | 34
  Immunologic Total; Week 52; n= 48, 104, 34 | 20.8 | 37.5 | 26.5
  Immunologic Total; Week 60; n= 48, 104, 34: number analyzed (Participants) | 48 | 104 | 34
  Immunologic Total; Week 60; n= 48, 104, 34 | 25.0 | 45.2 | 20.6
  Immunologic Total; Week 64; n= 48, 104, 34: number analyzed (Participants) | 48 | 104 | 34
  Immunologic Total; Week 64; n= 48, 104, 34 | 20.8 | 43.3 | 26.5
  Immunologic Total; Week 72; n=48, 104, 34: number analyzed (Participants) | 48 | 104 | 34
  Immunologic Total; Week 72; n=48, 104, 34 | 29.2 | 36.5 | 17.6
  Immunologic Total; Week 80; n=48, 104, 34: number analyzed (Participants) | 48 | 104 | 34
  Immunologic Total; Week 80; n=48, 104, 34 | 22.9 | 31.7 | 23.5
  Immunologic Total; Week 88; n=48, 104, 34: number analyzed (Participants) | 48 | 104 | 34
  Immunologic Total; Week 88; n=48, 104, 34 | 31.3 | 29.8 | 14.7
  Immunologic Total; Week 96; n=48, 104, 34: number analyzed (Participants) | 48 | 104 | 34
  Immunologic Total; Week 96; n=48, 104, 34 | 20.8 | 33.7 | 20.6
  Immunologic Total; Week 104; n=48, 104, 34: number analyzed (Participants) | 48 | 104 | 34
  Immunologic Total; Week 104; n=48, 104, 34 | 27.1 | 40.4 | 20.6
  Hematologic Total; Week 4; n= 8, 19, 3: number analyzed (Participants) | 8 | 19 | 3
  Hematologic Total; Week 4; n= 8, 19, 3 | 50.0 | 42.1 | 0
  Hematologic Total; Week 8; n= 8, 19, 3: number analyzed (Participants) | 8 | 19 | 3
  Hematologic Total; Week 8; n= 8, 19, 3 | 62.5 | 63.2 | 66.7
  Hematologic Total; Week 12; n= 8, 19, 3: number analyzed (Participants) | 8 | 19 | 3
  Hematologic Total; Week 12; n= 8, 19, 3 | 62.5 | 52.6 | 33.3
  Hematologic Total; Week 16; n= 8, 19, 3: number analyzed (Participants) | 8 | 19 | 3
  Hematologic Total; Week 16; n= 8, 19, 3 | 75.0 | 63.2 | 66.7
  Hematologic Total; Week 20; n= 8, 19, 3: number analyzed (Participants) | 8 | 19 | 3
  Hematologic Total; Week 20; n= 8, 19, 3 | 87.5 | 57.9 | 100
  Hematologic Total; Week 24; n= 8, 19, 3: number analyzed (Participants) | 8 | 19 | 3
  Hematologic Total; Week 24; n= 8, 19, 3 | 62.5 | 52.6 | 100
  Hematologic Total; Week 26; n= 8, 19, 3: number analyzed (Participants) | 8 | 19 | 3
  Hematologic Total; Week 26; n= 8, 19, 3 | 75.0 | 36.8 | 100
  Hematologic Total; Week 28; n= 8, 19, 3: number analyzed (Participants) | 8 | 19 | 3
  Hematologic Total; Week 28; n= 8, 19, 3 | 62.5 | 57.9 | 66.7
  Hematologic Total; Week 32; n= 8, 19, 3: number analyzed (Participants) | 8 | 19 | 3
  Hematologic Total; Week 32; n= 8, 19, 3 | 62.5 | 57.9 | 66.7
  Hematologic Total; Week 36; n= 8, 19, 3: number analyzed (Participants) | 8 | 19 | 3
  Hematologic Total; Week 36; n= 8, 19, 3 | 87.5 | 63.2 | 66.7
  Hematologic Total; Week 40; n= 8, 19, 3: number analyzed (Participants) | 8 | 19 | 3
  Hematologic Total; Week 40; n= 8, 19, 3 | 62.5 | 52.6 | 66.7
  Hematologic Total; Week 44; n= 8, 19, 3: number analyzed (Participants) | 8 | 19 | 3
  Hematologic Total; Week 44; n= 8, 19, 3 | 87.5 | 57.9 | 66.7
  Hematologic Total; Week 48; n= 8, 19, 3: number analyzed (Participants) | 8 | 19 | 3
  Hematologic Total; Week 48; n= 8, 19, 3 | 37.5 | 63.2 | 66.7
  Hematologic Total; Week 52; n= 8, 19, 3: number analyzed (Participants) | 8 | 19 | 3
  Hematologic Total; Week 52; n= 8, 19, 3 | 75.0 | 52.6 | 33.3
  Hematologic Total; Week 60; n= 8, 19, 3: number analyzed (Participants) | 8 | 19 | 3
  Hematologic Total; Week 60; n= 8, 19, 3 | 50.0 | 57.9 | 33.3
  Hematologic Total; Week 64; n= 8, 19, 3: number analyzed (Participants) | 8 | 19 | 3
  Hematologic Total; Week 64; n= 8, 19, 3 | 62.5 | 68.4 | 33.3
  Hematologic Total; Week 72; n= 8, 19, 3: number analyzed (Participants) | 8 | 19 | 3
  Hematologic Total; Week 72; n= 8, 19, 3 | 62.5 | 47.4 | 0
  Hematologic Total; Week 80; n= 8, 19, 3: number analyzed (Participants) | 8 | 19 | 3
  Hematologic Total; Week 80; n= 8, 19, 3 | 50.0 | 52.6 | 33.3
  Hematologic Total; Week 88; n= 8, 19, 3: number analyzed (Participants) | 8 | 19 | 3
  Hematologic Total; Week 88; n= 8, 19, 3 | 37.5 | 57.9 | 33.3
  Hematologic Total; Week 96; n= 8, 19, 3: number analyzed (Participants) | 8 | 19 | 3
  Hematologic Total; Week 96; n= 8, 19, 3 | 50.0 | 52.6 | 33.3
  Hematologic Total; Week 104; n= 8, 19, 3: number analyzed (Participants) | 8 | 19 | 3
  Hematologic Total; Week 104; n= 8, 19, 3 | 50.0 | 63.2 | 33.3

17. Secondary Outcome: Percentage of Participants With SLEDAI-2K Organ Worsening Compared to Baseline by Visits (PI Assessed)
Description: SLEDAI-2K assessments consisted of 24 individual items with 9 organ systems. Each item was given a weighted score(1 to 8 with higher score indicating increased activity)and summed if present at time of analysis. SLEDAI-2K score was sum of all 24 individual items from SLEDAI-2K, ranges from 0(no symptoms) to 105(presence of all defined symptoms). Higher scores indicates increased disease activity. A worsening was defined as an increase(compared to Baseline) in SLEDAI-2K score within same organ system at a post-Baseline visit. Baseline value was latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Percentage of participants with SLEDAI-2K organ worsening for following organ systems were reported;CNS total,Vascular total,Musculoskeletal total,Renal total,Mucocutaneous total,Cardio and Resp total,Immunologic total and Hematologic total. Constitutional organ system was removed from analysis and its one item (fever)moved to hematologic organ system.
Time Frame: Baseline (Day 1) and Weeks 4, 8, 12, 16, 20, 24, 26, 28, 32, 36, 40, 44, 48, 52, 60, 64, 72, 80, 88, 96, 104
Population: Modified Intent-to-Treat (MITT) Population. Only those participants with data available at specified time points were analyzed (represented by n=X in category titles). Only participants with no organ system involvement at Baseline were included.
Measure: Number; unit: Percentage of participants
Arm/Group | Belimumab + Placebo | Belimumab + Rituximab | Belimumab + Standard Therapy
Number analyzed (Participants) | 72 | 144 | 47
Percentage of participants
  CNS Total; Week 4; n= 69, 136, 43: number analyzed (Participants) | 69 | 136 | 43
  CNS Total; Week 4; n= 69, 136, 43 | 0 | 0 | 0
  CNS Total; Week 8; n= 64,132, 42: number analyzed (Participants) | 64 | 132 | 42
  CNS Total; Week 8; n= 64,132, 42 | 0 | 0 | 0
  CNS Total; Week 12; n= 65, 134, 42: number analyzed (Participants) | 65 | 134 | 42
  CNS Total; Week 12; n= 65, 134, 42 | 0 | 0 | 0
  CNS Total; Week 16; n= 65, 130, 42: number analyzed (Participants) | 65 | 130 | 42
  CNS Total; Week 16; n= 65, 130, 42 | 0 | 0.8 | 0
  CNS Total; Week 20; n= 63, 128, 42: number analyzed (Participants) | 63 | 128 | 42
  CNS Total; Week 20; n= 63, 128, 42 | 0 | 0 | 0
  CNS Total; Week 24; n= 61, 127, 41: number analyzed (Participants) | 61 | 127 | 41
  CNS Total; Week 24; n= 61, 127, 41 | 0 | 0.8 | 0
  CNS Total; Week 26; n=61, 116, 38: number analyzed (Participants) | 61 | 116 | 38
  CNS Total; Week 26; n=61, 116, 38 | 0 | 0.9 | 0
  CNS Total; Week 28; n=62, 124, 41: number analyzed (Participants) | 62 | 124 | 41
  CNS Total; Week 28; n=62, 124, 41 | 0 | 0 | 0
  CNS Total; Week 32; n= 61, 124, 41: number analyzed (Participants) | 61 | 124 | 41
  CNS Total; Week 32; n= 61, 124, 41 | 0 | 0.8 | 0
  CNS Total; Week 36; n=61, 124, 41: number analyzed (Participants) | 61 | 124 | 41
  CNS Total; Week 36; n=61, 124, 41 | 0 | 1.6 | 0
  CNS Total; Week 40; n=61, 123, 41: number analyzed (Participants) | 61 | 123 | 41
  CNS Total; Week 40; n=61, 123, 41 | 0 | 0 | 0
  CNS Total; Week 44; n= 61, 121, 41: number analyzed (Participants) | 61 | 121 | 41
  CNS Total; Week 44; n= 61, 121, 41 | 0 | 0 | 0
  CNS Total; Week 48; n= 58, 120,39: number analyzed (Participants) | 58 | 120 | 39
  CNS Total; Week 48; n= 58, 120,39 | 0 | 0 | 0
  CNS Total; Week 52; n= 62, 120, 38: number analyzed (Participants) | 62 | 120 | 38
  CNS Total; Week 52; n= 62, 120, 38 | 0 | 0 | 0
  CNS Total; Week 60; n=59, 117, 35: number analyzed (Participants) | 59 | 117 | 35
  CNS Total; Week 60; n=59, 117, 35 | 0 | 0 | 0
  CNS Total; Week 64; n=60, 117, 34: number analyzed (Participants) | 60 | 117 | 34
  CNS Total; Week 64; n=60, 117, 34 | 0 | 0 | 0
  CNS Total; Week 72; n= 56, 109, 31: number analyzed (Participants) | 56 | 109 | 31
  CNS Total; Week 72; n= 56, 109, 31 | 0 | 0 | 0
  CNS Total; Week 80; n=55, 111, 35: number analyzed (Participants) | 55 | 111 | 35
  CNS Total; Week 80; n=55, 111, 35 | 0 | 0 | 0
  CNS Total; Week 88; n= 57, 107, 34: number analyzed (Participants) | 57 | 107 | 34
  CNS Total; Week 88; n= 57, 107, 34 | 0 | 0 | 0
  CNS Total; Week 96; n=52, 107, 33: number analyzed (Participants) | 52 | 107 | 33
  CNS Total; Week 96; n=52, 107, 33 | 0 | 0 | 0
  CNS Total; Week 104; n= 53, 112, 34: number analyzed (Participants) | 53 | 112 | 34
  CNS Total; Week 104; n= 53, 112, 34 | 0 | 0 | 0
  Vascular Total;Week 4; n= 65, 128, 45: number analyzed (Participants) | 65 | 128 | 45
  Vascular Total;Week 4; n= 65, 128, 45 | 0 | 3.9 | 0
  Vascular Total;Week 8; n= 61, 124, 44: number analyzed (Participants) | 61 | 124 | 44
  Vascular Total;Week 8; n= 61, 124, 44 | 0 | 2.4 | 0
  Vascular Total; Week 12; n= 62, 126, 44: number analyzed (Participants) | 62 | 126 | 44
  Vascular Total; Week 12; n= 62, 126, 44 | 1.6 | 1.6 | 0
  Vascular Total; Week 16; n=62, 122, 44: number analyzed (Participants) | 62 | 122 | 44
  Vascular Total; Week 16; n=62, 122, 44 | 0 | 1.6 | 0
  Vascular Total; Week 20; n=60, 120, 44: number analyzed (Participants) | 60 | 120 | 44
  Vascular Total; Week 20; n=60, 120, 44 | 0 | 0.8 | 0
  Vascular Total; Week 24; n= 59, 119, 43: number analyzed (Participants) | 59 | 119 | 43
  Vascular Total; Week 24; n= 59, 119, 43 | 0 | 0 | 0
  Vascular Total; Week 26; n=58, 109, 40: number analyzed (Participants) | 58 | 109 | 40
  Vascular Total; Week 26; n=58, 109, 40 | 0 | 0.9 | 0
  Vascular Total;Week 28; n= 61, 116, 43: number analyzed (Participants) | 61 | 116 | 43
  Vascular Total;Week 28; n= 61, 116, 43 | 0 | 1.7 | 0
  Vascular Total;Week 32; n=59, 116, 43: number analyzed (Participants) | 59 | 116 | 43
  Vascular Total;Week 32; n=59, 116, 43 | 0 | 2.6 | 0
  Vascular Total;Week 36; n= 59, 116, 43: number analyzed (Participants) | 59 | 116 | 43
  Vascular Total;Week 36; n= 59, 116, 43 | 0 | 1.7 | 0
  Vascular Total;Week 40; n=59, 115, 43: number analyzed (Participants) | 59 | 115 | 43
  Vascular Total;Week 40; n=59, 115, 43 | 0 | 1.7 | 0
  Vascular Total;Week 44; n= 59, 113, 43: number analyzed (Participants) | 59 | 113 | 43
  Vascular Total;Week 44; n= 59, 113, 43 | 0 | 0 | 0
  Vascular Total;Week 48; n= 57, 112, 40: number analyzed (Participants) | 57 | 112 | 40
  Vascular Total;Week 48; n= 57, 112, 40 | 0 | 0 | 0
  Vascular Total;Week 52; n=60, 112, 40: number analyzed (Participants) | 60 | 112 | 40
  Vascular Total;Week 52; n=60, 112, 40 | 0 | 0.9 | 0
  Vascular Total;Week 60; n= 58, 109, 37: number analyzed (Participants) | 58 | 109 | 37
  Vascular Total;Week 60; n= 58, 109, 37 | 0 | 0 | 0
  Vascular Total;Week 64; n=59, 109, 36: number analyzed (Participants) | 59 | 109 | 36
  Vascular Total;Week 64; n=59, 109, 36 | 0 | 1.8 | 0
  Vascular Total;Week 72; n=55, 101, 33: number analyzed (Participants) | 55 | 101 | 33
  Vascular Total;Week 72; n=55, 101, 33 | 0 | 0 | 0
  Vascular Total;Week 80; n= 54, 104, 37: number analyzed (Participants) | 54 | 104 | 37
  Vascular Total;Week 80; n= 54, 104, 37 | 0 | 1.0 | 0
  Vascular Total;Week 88; n=56, 102, 36: number analyzed (Participants) | 56 | 102 | 36
  Vascular Total;Week 88; n=56, 102, 36 | 0 | 0 | 0
  Vascular Total;Week 96; n=51, 101, 35: number analyzed (Participants) | 51 | 101 | 35
  Vascular Total;Week 96; n=51, 101, 35 | 0 | 0 | 0
  Vascular Total;Week 104; n=53, 105, 36: number analyzed (Participants) | 53 | 105 | 36
  Vascular Total;Week 104; n=53, 105, 36 | 0 | 0 | 0
  Musculoskeletal Total; Week 4; n=15, 33, 12: number analyzed (Participants) | 15 | 33 | 12
  Musculoskeletal Total; Week 4; n=15, 33, 12 | 0 | 12.1 | 0
  Musculoskeletal Total; Week 8; n= 15, 33, 12: number analyzed (Participants) | 15 | 33 | 12
  Musculoskeletal Total; Week 8; n= 15, 33, 12 | 6.7 | 6.1 | 0
  Musculoskeletal Total; Week 12; n= 15, 33, 12: number analyzed (Participants) | 15 | 33 | 12
  Musculoskeletal Total; Week 12; n= 15, 33, 12 | 13.3 | 6.1 | 0
  Musculoskeletal Total; Week 16; n= 15, 32, 12: number analyzed (Participants) | 15 | 32 | 12
  Musculoskeletal Total; Week 16; n= 15, 32, 12 | 6.7 | 3.1 | 8.3
  Musculoskeletal Total; Week 20; n= 15, 32, 12: number analyzed (Participants) | 15 | 32 | 12
  Musculoskeletal Total; Week 20; n= 15, 32, 12 | 6.7 | 6.3 | 0
  Musculoskeletal Total; Week 24; n= 15, 31, 11: number analyzed (Participants) | 15 | 31 | 11
  Musculoskeletal Total; Week 24; n= 15, 31, 11 | 0 | 6.5 | 0
  Musculoskeletal Total; Week 26; n= 15, 31, 11: number analyzed (Participants) | 15 | 31 | 11
  Musculoskeletal Total; Week 26; n= 15, 31, 11 | 0 | 3.2 | 0
  Musculoskeletal Total; Week 28; n= 14, 31, 11: number analyzed (Participants) | 14 | 31 | 11
  Musculoskeletal Total; Week 28; n= 14, 31, 11 | 0 | 3.2 | 9.1
  Musculoskeletal Total; Week 32; n= 15, 30, 11: number analyzed (Participants) | 15 | 30 | 11
  Musculoskeletal Total; Week 32; n= 15, 30, 11 | 0 | 6.7 | 9.1
  Musculoskeletal Total; Week 36; n= 14, 30, 11: number analyzed (Participants) | 14 | 30 | 11
  Musculoskeletal Total; Week 36; n= 14, 30, 11 | 7.1 | 3.3 | 9.1
  Musculoskeletal Total; Week 40; n=15, 30, 11: number analyzed (Participants) | 15 | 30 | 11
  Musculoskeletal Total; Week 40; n=15, 30, 11 | 0 | 3.3 | 9.1
  Musculoskeletal Total; Week 44; n=15, 29, 11: number analyzed (Participants) | 15 | 29 | 11
  Musculoskeletal Total; Week 44; n=15, 29, 11 | 0 | 6.9 | 9.1
  Musculoskeletal Total; Week 48; n= 14, 30, 10: number analyzed (Participants) | 14 | 30 | 10
  Musculoskeletal Total; Week 48; n= 14, 30, 10 | 7.1 | 3.3 | 10.0
  Musculoskeletal Total; Week 52; n= 15, 30, 11: number analyzed (Participants) | 15 | 30 | 11
  Musculoskeletal Total; Week 52; n= 15, 30, 11 | 6.7 | 6.7 | 9.1
  Musculoskeletal Total; Week 60; n= 14, 28, 11: number analyzed (Participants) | 14 | 28 | 11
  Musculoskeletal Total; Week 60; n= 14, 28, 11 | 0 | 0 | 9.1
  Musculoskeletal Total; Week 64; n=14, 29, 10: number analyzed (Participants) | 14 | 29 | 10
  Musculoskeletal Total; Week 64; n=14, 29, 10 | 0 | 3.4 | 10.0
  Musculoskeletal Total; Week 72; n= 14, 27, 10: number analyzed (Participants) | 14 | 27 | 10
  Musculoskeletal Total; Week 72; n= 14, 27, 10 | 0 | 11.1 | 10.0
  Musculoskeletal Total; Week 80; n= 13, 26, 9: number analyzed (Participants) | 13 | 26 | 9
  Musculoskeletal Total; Week 80; n= 13, 26, 9 | 0 | 0 | 11.1
  Musculoskeletal Total; Week 88; n= 13, 25, 9: number analyzed (Participants) | 13 | 25 | 9
  Musculoskeletal Total; Week 88; n= 13, 25, 9 | 15.4 | 4.0 | 0
  Musculoskeletal Total; Week 96; n= 12, 26, 9: number analyzed (Participants) | 12 | 26 | 9
  Musculoskeletal Total; Week 96; n= 12, 26, 9 | 0 | 3.8 | 0
  Musculoskeletal Total; Week 104; n= 13, 27, 9: number analyzed (Participants) | 13 | 27 | 9
  Musculoskeletal Total; Week 104; n= 13, 27, 9 | 0 | 0 | 0
  Renal Total; Week 4; n= 57, 117, 36: number analyzed (Participants) | 57 | 117 | 36
  Renal Total; Week 4; n= 57, 117, 36 | 5.3 | 6.0 | 11.1
  Renal Total; Week 8; n=51, 110, 36: number analyzed (Participants) | 51 | 110 | 36
  Renal Total; Week 8; n=51, 110, 36 | 2.0 | 3.6 | 5.6
  Renal Total; Week 12; n=53, 115, 35: number analyzed (Participants) | 53 | 115 | 35
  Renal Total; Week 12; n=53, 115, 35 | 1.9 | 3.5 | 8.6
  Renal Total; Week 16; n=53, 112, 35: number analyzed (Participants) | 53 | 112 | 35
  Renal Total; Week 16; n=53, 112, 35 | 7.5 | 4.5 | 2.9
  Renal Total; Week 20; n= 49, 108, 36: number analyzed (Participants) | 49 | 108 | 36
  Renal Total; Week 20; n= 49, 108, 36 | 8.2 | 3.7 | 8.3
  Renal Total; Week 24; n= 49, 111, 35: number analyzed (Participants) | 49 | 111 | 35
  Renal Total; Week 24; n= 49, 111, 35 | 10.2 | 3.6 | 2.9
  Renal Total; Week 26; n= 49, 99, 33: number analyzed (Participants) | 49 | 99 | 33
  Renal Total; Week 26; n= 49, 99, 33 | 6.1 | 0 | 0
  Renal Total; Week 28; n= 50, 106, 36: number analyzed (Participants) | 50 | 106 | 36
  Renal Total; Week 28; n= 50, 106, 36 | 10.0 | 1.9 | 2.8
  Renal Total; Week 32; n= 50,107, 36: number analyzed (Participants) | 50 | 107 | 36
  Renal Total; Week 32; n= 50,107, 36 | 6.0 | 2.8 | 2.8
  Renal Total; Week 36; n= 50, 107, 36: number analyzed (Participants) | 50 | 107 | 36
  Renal Total; Week 36; n= 50, 107, 36 | 8.0 | 2.8 | 5.6
  Renal Total; Week 40; n= 47, 106, 34: number analyzed (Participants) | 47 | 106 | 34
  Renal Total; Week 40; n= 47, 106, 34 | 6.4 | 4.7 | 0
  Renal Total; Week 44; n= 49, 103, 35: number analyzed (Participants) | 49 | 103 | 35
  Renal Total; Week 44; n= 49, 103, 35 | 6.1 | 1.0 | 2.9
  Renal Total; Week 48; n= 47, 101, 32: number analyzed (Participants) | 47 | 101 | 32
  Renal Total; Week 48; n= 47, 101, 32 | 10.6 | 5.9 | 6.3
  Renal Total; Week 52; n= 49, 103, 32: number analyzed (Participants) | 49 | 103 | 32
  Renal Total; Week 52; n= 49, 103, 32 | 8.2 | 3.9 | 3.1
  Renal Total; Week 60; n=47, 96, 30: number analyzed (Participants) | 47 | 96 | 30
  Renal Total; Week 60; n=47, 96, 30 | 6.4 | 4.2 | 0
  Renal Total; Week 64; n= 50, 99, 29: number analyzed (Participants) | 50 | 99 | 29
  Renal Total; Week 64; n= 50, 99, 29 | 2.0 | 2.0 | 0
  Renal Total; Week 72; n= 40, 89, 26: number analyzed (Participants) | 40 | 89 | 26
  Renal Total; Week 72; n= 40, 89, 26 | 5.0 | 4.5 | 0
  Renal Total; Week 80; n= 41, 90, 29: number analyzed (Participants) | 41 | 90 | 29
  Renal Total; Week 80; n= 41, 90, 29 | 14.6 | 3.3 | 6.9
  Renal Total; Week 88; n= 44, 85, 29: number analyzed (Participants) | 44 | 85 | 29
  Renal Total; Week 88; n= 44, 85, 29 | 13.6 | 1.2 | 0
  Renal Total; Week 96; n= 43, 85, 29: number analyzed (Participants) | 43 | 85 | 29
  Renal Total; Week 96; n= 43, 85, 29 | 4.7 | 1.2 | 0
  Renal Total; Week 104; n= 44, 90, 30: number analyzed (Participants) | 44 | 90 | 30
  Renal Total; Week 104; n= 44, 90, 30 | 6.8 | 2.2 | 0
  Mucocutaneous Total; Week 4; n= 13, 18, 4: number analyzed (Participants) | 13 | 18 | 4
  Mucocutaneous Total; Week 4; n= 13, 18, 4 | 15.4 | 5.6 | 0
  Mucocutaneous Total; Week 8; n= 12, 18, 4: number analyzed (Participants) | 12 | 18 | 4
  Mucocutaneous Total; Week 8; n= 12, 18, 4 | 8.3 | 11.1 | 0
  Mucocutaneous Total; Week 12; n= 12, 18, 4: number analyzed (Participants) | 12 | 18 | 4
  Mucocutaneous Total; Week 12; n= 12, 18, 4 | 8.3 | 16.7 | 0
  Mucocutaneous Total; Week 16; n= 12, 18, 4: number analyzed (Participants) | 12 | 18 | 4
  Mucocutaneous Total; Week 16; n= 12, 18, 4 | 0 | 5.6 | 0
  Mucocutaneous Total; Week 20; n= 12, 18, 4: number analyzed (Participants) | 12 | 18 | 4
  Mucocutaneous Total; Week 20; n= 12, 18, 4 | 25.0 | 5.6 | 0
  Mucocutaneous Total; Week 24; n= 11, 17, 4: number analyzed (Participants) | 11 | 17 | 4
  Mucocutaneous Total; Week 24; n= 11, 17, 4 | 18.2 | 5.9 | 0
  Mucocutaneous Total; Week 26; n= 10, 17, 4: number analyzed (Participants) | 10 | 17 | 4
  Mucocutaneous Total; Week 26; n= 10, 17, 4 | 20.0 | 11.8 | 0
  Mucocutaneous Total; Week 28; n= 10, 17, 4: number analyzed (Participants) | 10 | 17 | 4
  Mucocutaneous Total; Week 28; n= 10, 17, 4 | 0 | 11.8 | 0
  Mucocutaneous Total; Week 32; n= 10, 17, 4: number analyzed (Participants) | 10 | 17 | 4
  Mucocutaneous Total; Week 32; n= 10, 17, 4 | 10.0 | 5.9 | 0
  Mucocutaneous Total; Week 36; n= 10, 17, 4: number analyzed (Participants) | 10 | 17 | 4
  Mucocutaneous Total; Week 36; n= 10, 17, 4 | 0 | 5.9 | 0
  Mucocutaneous Total; Week 40; n= 10, 17, 4: number analyzed (Participants) | 10 | 17 | 4
  Mucocutaneous Total; Week 40; n= 10, 17, 4 | 20.0 | 11.8 | 0
  Mucocutaneous Total; Week 44; n= 10, 17, 4: number analyzed (Participants) | 10 | 17 | 4
  Mucocutaneous Total; Week 44; n= 10, 17, 4 | 10.0 | 0 | 0
  Mucocutaneous Total; Week 48; n=10, 16, 3: number analyzed (Participants) | 10 | 16 | 3
  Mucocutaneous Total; Week 48; n=10, 16, 3 | 0 | 6.3 | 0
  Mucocutaneous Total; Week 52; n= 10, 17, 4: number analyzed (Participants) | 10 | 17 | 4
  Mucocutaneous Total; Week 52; n= 10, 17, 4 | 0 | 5.9 | 25.0
  Mucocutaneous Total; Week 60; n= 9, 17, 4: number analyzed (Participants) | 9 | 17 | 4
  Mucocutaneous Total; Week 60; n= 9, 17, 4 | 11.1 | 11.8 | 0
  Mucocutaneous Total; Week 64; n= 10, 16, 4: number analyzed (Participants) | 10 | 16 | 4
  Mucocutaneous Total; Week 64; n= 10, 16, 4 | 0 | 6.3 | 25.0
  Mucocutaneous Total; Week 72; n=10, 16, 4: number analyzed (Participants) | 10 | 16 | 4
  Mucocutaneous Total; Week 72; n=10, 16, 4 | 20 | 6.3 | 25.0
  Mucocutaneous Total; Week 80; n= 9, 17, 4: number analyzed (Participants) | 9 | 17 | 4
  Mucocutaneous Total; Week 80; n= 9, 17, 4 | 0 | 0 | 25.0
  Mucocutaneous Total; Week 88; n= 9, 16, 4: number analyzed (Participants) | 9 | 16 | 4
  Mucocutaneous Total; Week 88; n= 9, 16, 4 | 0 | 6.3 | 25.0
  Mucocutaneous Total; Week 96; n= 9, 15, 4: number analyzed (Participants) | 9 | 15 | 4
  Mucocutaneous Total; Week 96; n= 9, 15, 4 | 11.1 | 0 | 25.0
  Mucocutaneous Total; Week 104; n= 9, 17, 4: number analyzed (Participants) | 9 | 17 | 4
  Mucocutaneous Total; Week 104; n= 9, 17, 4 | 11.1 | 5.9 | 0
  Cardio and Resp Total; Week 4; n= 68, 132, 45: number analyzed (Participants) | 68 | 132 | 45
  Cardio and Resp Total; Week 4; n= 68, 132, 45 | 2.9 | 0.8 | 0
  Cardio and Resp Total; Week 8; n= 63, 128, 44: number analyzed (Participants) | 63 | 128 | 44
  Cardio and Resp Total; Week 8; n= 63, 128, 44 | 0 | 0.8 | 0
  Cardio and Resp Total; Week 12; n= 64, 130, 44: number analyzed (Participants) | 64 | 130 | 44
  Cardio and Resp Total; Week 12; n= 64, 130, 44 | 0 | 0.8 | 0
  Cardio and Resp Total; Week 16; n= 64, 126, 44: number analyzed (Participants) | 64 | 126 | 44
  Cardio and Resp Total; Week 16; n= 64, 126, 44 | 3.1 | 0 | 0
  Cardio and Resp Total; Week 20; n= 63, 124, 44: number analyzed (Participants) | 63 | 124 | 44
  Cardio and Resp Total; Week 20; n= 63, 124, 44 | 1.6 | 0.8 | 0
  Cardio and Resp Total; Week 24; n= 60, 123, 43: number analyzed (Participants) | 60 | 123 | 43
  Cardio and Resp Total; Week 24; n= 60, 123, 43 | 0 | 0 | 0
  Cardio and Resp Total; Week 26; n=59, 112, 40: number analyzed (Participants) | 59 | 112 | 40
  Cardio and Resp Total; Week 26; n=59, 112, 40 | 0 | 0 | 0
  Cardio and Resp Total; Week 28; n= 61, 120, 43: number analyzed (Participants) | 61 | 120 | 43
  Cardio and Resp Total; Week 28; n= 61, 120, 43 | 3.3 | 0.8 | 0
  Cardio and Resp Total; Week 32; n= 60, 120, 43: number analyzed (Participants) | 60 | 120 | 43
  Cardio and Resp Total; Week 32; n= 60, 120, 43 | 1.7 | 0 | 0
  Cardio and Resp Total; Week 36; n= 60, 120, 43: number analyzed (Participants) | 60 | 120 | 43
  Cardio and Resp Total; Week 36; n= 60, 120, 43 | 1.7 | 0 | 0
  Cardio and Resp Total; Week 40; n=60, 119, 43: number analyzed (Participants) | 60 | 119 | 43
  Cardio and Resp Total; Week 40; n=60, 119, 43 | 0 | 0 | 0
  Cardio and Resp Total; Week 44; n= 60, 117, 43: number analyzed (Participants) | 60 | 117 | 43
  Cardio and Resp Total; Week 44; n= 60, 117, 43 | 1.7 | 0 | 0
  Cardio and Resp Total; Week 48; n= 57, 116, 40: number analyzed (Participants) | 57 | 116 | 40
  Cardio and Resp Total; Week 48; n= 57, 116, 40 | 0 | 0 | 2.5
  Cardio and Resp Total; Week 52; n=61, 116, 40: number analyzed (Participants) | 61 | 116 | 40
  Cardio and Resp Total; Week 52; n=61, 116, 40 | 0 | 0 | 0
  Cardio and Resp Total; Week 60; n= 58, 114, 37: number analyzed (Participants) | 58 | 114 | 37
  Cardio and Resp Total; Week 60; n= 58, 114, 37 | 0 | 0 | 0
  Cardio and Resp Total; Week 64; n= 59, 114, 36: number analyzed (Participants) | 59 | 114 | 36
  Cardio and Resp Total; Week 64; n= 59, 114, 36 | 0 | 0.9 | 0
  Cardio and Resp Total; Week 72; n= 55, 106, 33: number analyzed (Participants) | 55 | 106 | 33
  Cardio and Resp Total; Week 72; n= 55, 106, 33 | 0 | 0 | 0
  Cardio and Resp Total; Week 80; n= 54, 107, 37: number analyzed (Participants) | 54 | 107 | 37
  Cardio and Resp Total; Week 80; n= 54, 107, 37 | 1.9 | 0 | 0
  Cardio and Resp Total; Week 88; n= 56, 104, 36: number analyzed (Participants) | 56 | 104 | 36
  Cardio and Resp Total; Week 88; n= 56, 104, 36 | 1.8 | 0 | 0
  Cardio and Resp Total; Week 96; n=51, 104, 35: number analyzed (Participants) | 51 | 104 | 35
  Cardio and Resp Total; Week 96; n=51, 104, 35 | 0 | 1.0 | 0
  Cardio and Resp Total; Week 104; n= 52, 109, 36: number analyzed (Participants) | 52 | 109 | 36
  Cardio and Resp Total; Week 104; n= 52, 109, 36 | 0 | 0 | 0
  Immunologic Total; Week 4; n=23, 37, 13: number analyzed (Participants) | 23 | 37 | 13
  Immunologic Total; Week 4; n=23, 37, 13 | 17.4 | 0 | 7.7
  Immunologic Total; Week 8; n=20, 37, 12: number analyzed (Participants) | 20 | 37 | 12
  Immunologic Total; Week 8; n=20, 37, 12 | 20.0 | 10.8 | 0
  Immunologic Total; Week 12; n=21, 37,12: number analyzed (Participants) | 21 | 37 | 12
  Immunologic Total; Week 12; n=21, 37,12 | 23.8 | 8.1 | 16.7
  Immunologic Total; Week 16; n= 21, 35, 12: number analyzed (Participants) | 21 | 35 | 12
  Immunologic Total; Week 16; n= 21, 35, 12 | 9.5 | 11.4 | 0
  Immunologic Total; Week 20; n= 19, 35, 12: number analyzed (Participants) | 19 | 35 | 12
  Immunologic Total; Week 20; n= 19, 35, 12 | 15.8 | 11.4 | 0
  Immunologic Total; Week 24; n= 18, 35, 12: number analyzed (Participants) | 18 | 35 | 12
  Immunologic Total; Week 24; n= 18, 35, 12 | 5.6 | 5.7 | 0
  Immunologic Total; Week 26; n= 18, 30, 12: number analyzed (Participants) | 18 | 30 | 12
  Immunologic Total; Week 26; n= 18, 30, 12 | 5.6 | 6.7 | 8.3
  Immunologic Total; Week 28; n= 19, 35, 12: number analyzed (Participants) | 19 | 35 | 12
  Immunologic Total; Week 28; n= 19, 35, 12 | 15.8 | 8.6 | 16.7
  Immunologic Total; Week 32; n= 19, 33, 12: number analyzed (Participants) | 19 | 33 | 12
  Immunologic Total; Week 32; n= 19, 33, 12 | 10.5 | 12.1 | 8.3
  Immunologic Total; Week 36; n= 19, 34, 12: number analyzed (Participants) | 19 | 34 | 12
  Immunologic Total; Week 36; n= 19, 34, 12 | 15.8 | 8.8 | 16.7
  Immunologic Total; Week 40; n= 19, 33, 12: number analyzed (Participants) | 19 | 33 | 12
  Immunologic Total; Week 40; n= 19, 33, 12 | 21.1 | 6.1 | 8.3
  Immunologic Total; Week 44; n= 18, 33, 12: number analyzed (Participants) | 18 | 33 | 12
  Immunologic Total; Week 44; n= 18, 33, 12 | 22.2 | 0 | 0
  Immunologic Total; Week 48; n= 18, 33, 11: number analyzed (Participants) | 18 | 33 | 11
  Immunologic Total; Week 48; n= 18, 33, 11 | 22.2 | 3.0 | 27.3
  Immunologic Total; Week 52; n= 19, 32, 12: number analyzed (Participants) | 19 | 32 | 12
  Immunologic Total; Week 52; n= 19, 32, 12 | 21.1 | 3.1 | 8.3
  Immunologic Total; Week 60; n= 18, 32, 10: number analyzed (Participants) | 18 | 32 | 10
  Immunologic Total; Week 60; n= 18, 32, 10 | 16.7 | 6.3 | 0
  Immunologic Total; Week 64; n= 19, 33, 10: number analyzed (Participants) | 19 | 33 | 10
  Immunologic Total; Week 64; n= 19, 33, 10 | 21.1 | 6.1 | 20.0
  Immunologic Total; Week 72; n= 17, 28, 9: number analyzed (Participants) | 17 | 28 | 9
  Immunologic Total; Week 72; n= 17, 28, 9 | 23.5 | 7.1 | 11.1
  Immunologic Total; Week 80; n= 18, 29, 11: number analyzed (Participants) | 18 | 29 | 11
  Immunologic Total; Week 80; n= 18, 29, 11 | 5.6 | 6.9 | 18.2
  Immunologic Total; Week 88; n= 19, 29, 11: number analyzed (Participants) | 19 | 29 | 11
  Immunologic Total; Week 88; n= 19, 29, 11 | 10.5 | 6.9 | 18.2
  Immunologic Total; Week 96; n= 16, 30, 11: number analyzed (Participants) | 16 | 30 | 11
  Immunologic Total; Week 96; n= 16, 30, 11 | 12.5 | 13.3 | 18.2
  Immunologic Total; Week 104; n= 17, 28, 12: number analyzed (Participants) | 17 | 28 | 12
  Immunologic Total; Week 104; n= 17, 28, 12 | 11.8 | 17.9 | 16.7
  Hematologic Total; Week 4; n= 59, 115, 40: number analyzed (Participants) | 59 | 115 | 40
  Hematologic Total; Week 4; n= 59, 115, 40 | 5.1 | 3.5 | 5.0
  Hematologic Total; Week 8; n= 52, 109, 38: number analyzed (Participants) | 52 | 109 | 38
  Hematologic Total; Week 8; n= 52, 109, 38 | 3.8 | 5.5 | 0
  Hematologic Total; Week 12; n= 55, 110, 38: number analyzed (Participants) | 55 | 110 | 38
  Hematologic Total; Week 12; n= 55, 110, 38 | 1.8 | 4.5 | 10.5
  Hematologic Total; Week 16; n=54, 107, 34: number analyzed (Participants) | 54 | 107 | 34
  Hematologic Total; Week 16; n=54, 107, 34 | 1.9 | 2.8 | 2.9
  Hematologic Total; Week 20; n= 54, 108, 40: number analyzed (Participants) | 54 | 108 | 40
  Hematologic Total; Week 20; n= 54, 108, 40 | 5.6 | 5.6 | 5.0
  Hematologic Total; Week 24; n= 53, 111, 37: number analyzed (Participants) | 53 | 111 | 37
  Hematologic Total; Week 24; n= 53, 111, 37 | 3.8 | 2.7 | 2.7
  Hematologic Total; Week 26; n= 53, 101, 37: number analyzed (Participants) | 53 | 101 | 37
  Hematologic Total; Week 26; n= 53, 101, 37 | 9.4 | 5.0 | 10.8
  Hematologic Total; Week 28; n= 52, 106, 39: number analyzed (Participants) | 52 | 106 | 39
  Hematologic Total; Week 28; n= 52, 106, 39 | 7.7 | 3.8 | 5.1
  Hematologic Total; Week 32; n=52, 110, 38: number analyzed (Participants) | 52 | 110 | 38
  Hematologic Total; Week 32; n=52, 110, 38 | 0 | 4.5 | 7.9
  Hematologic Total; Week 36; n= 53, 109, 40: number analyzed (Participants) | 53 | 109 | 40
  Hematologic Total; Week 36; n= 53, 109, 40 | 5.7 | 6.4 | 2.5
  Hematologic Total; Week 40; n= 51, 108, 37: number analyzed (Participants) | 51 | 108 | 37
  Hematologic Total; Week 40; n= 51, 108, 37 | 0 | 10.2 | 5.4
  Hematologic Total; Week 44; n=53, 107, 38: number analyzed (Participants) | 53 | 107 | 38
  Hematologic Total; Week 44; n=53, 107, 38 | 7.5 | 6.5 | 5.3
  Hematologic Total; Week 48; n=51, 105, 35: number analyzed (Participants) | 51 | 105 | 35
  Hematologic Total; Week 48; n=51, 105, 35 | 5.9 | 4.8 | 0
  Hematologic Total; Week 52; n= 53, 103, 37: number analyzed (Participants) | 53 | 103 | 37
  Hematologic Total; Week 52; n= 53, 103, 37 | 3.8 | 3.9 | 2.7
  Hematologic Total; Week 60; n=53, 101, 35: number analyzed (Participants) | 53 | 101 | 35
  Hematologic Total; Week 60; n=53, 101, 35 | 9.4 | 5.0 | 5.7
  Hematologic Total; Week 64; n=54, 98, 32: number analyzed (Participants) | 54 | 98 | 32
  Hematologic Total; Week 64; n=54, 98, 32 | 11.1 | 5.1 | 6.3
  Hematologic Total; Week 72; n= 47,96, 29: number analyzed (Participants) | 47 | 96 | 29
  Hematologic Total; Week 72; n= 47,96, 29 | 10.6 | 5.2 | 3.4
  Hematologic Total; Week 80; n= 45, 94, 35: number analyzed (Participants) | 45 | 94 | 35
  Hematologic Total; Week 80; n= 45, 94, 35 | 0 | 4.3 | 5.7
  Hematologic Total; Week 88; n= 46, 88, 32: number analyzed (Participants) | 46 | 88 | 32
  Hematologic Total; Week 88; n= 46, 88, 32 | 10.9 | 9.1 | 3.1
  Hematologic Total; Week 96; n= 45, 90, 32: number analyzed (Participants) | 45 | 90 | 32
  Hematologic Total; Week 96; n= 45, 90, 32 | 4.4 | 4.4 | 3.1
  Hematologic Total; Week 104; n= 46, 94, 32: number analyzed (Participants) | 46 | 94 | 32
  Hematologic Total; Week 104; n= 46, 94, 32 | 4.3 | 6.4 | 6.3

18. Secondary Outcome: Change From Baseline in Physician Global Assessment (PGA) by Visits
Description: The Physician's Global Assessment (PGA) was a physician-reported visual analogue scale that provides an overall measure of the participant's current disease activity. Physician's Global Assessment was collected on a 10 centimeter (cm) visual analogue scale (VAS) by placing a mark on the scale between 0 (no disease activity) to 10 (maximum disease activity). The PGA score was then rescaled for reporting by multiplying the collected score by 3 divided by 10. Hence, the PGA score ranges from 0 to 3 with higher scores indicating greater disease activity. Baseline value was the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was defined as the post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1) and Weeks 4, 8, 12, 16, 20, 24, 26, 28, 32, 36, 40, 44, 48, 52, 60, 64, 72, 80, 88, 96, 104
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Belimumab + Placebo | Belimumab + Rituximab | Belimumab + Standard Therapy
Number analyzed (Participants) | 72 | 144 | 47
Scores on a scale
  Week 4; n=72, 142, 45: number analyzed (Participants) | 72 | 142 | 45
  Week 4; n=72, 142, 45 | -0.285 (0.4816) | -0.247 (0.4640) | -0.303 (0.5464)
  Week 8; n=66, 135, 44: number analyzed (Participants) | 66 | 135 | 44
  Week 8; n=66, 135, 44 | -0.535 (0.5134) | -0.520 (0.5243) | -0.585 (0.5793)
  Week 12; n=66, 137, 44: number analyzed (Participants) | 66 | 137 | 44
  Week 12; n=66, 137, 44 | -0.592 (0.5265) | -0.660 (0.5776) | -0.654 (0.5450)
  Week 16; n=68, 132, 44: number analyzed (Participants) | 68 | 132 | 44
  Week 16; n=68, 132, 44 | -0.619 (0.5475) | -0.717 (0.5802) | -0.759 (0.6072)
  Week 20; n=66, 130, 44: number analyzed (Participants) | 66 | 130 | 44
  Week 20; n=66, 130, 44 | -0.697 (0.6157) | -0.787 (0.5445) | -0.786 (0.6772)
  Week 24; n=62, 130, 43: number analyzed (Participants) | 62 | 130 | 43
  Week 24; n=62, 130, 43 | -0.770 (0.5888) | -0.766 (0.5059) | -0.965 (0.6413)
  Week 26; n=62, 120, 40: number analyzed (Participants) | 62 | 120 | 40
  Week 26; n=62, 120, 40 | -0.786 (0.5727) | -0.811 (0.5445) | -0.929 (0.6631)
  Week 28; n=63, 127, 43: number analyzed (Participants) | 63 | 127 | 43
  Week 28; n=63, 127, 43 | -0.781 (0.5395) | -0.817 (0.5360) | -0.980 (0.6286)
  Week 32; n=62, 124, 43: number analyzed (Participants) | 62 | 124 | 43
  Week 32; n=62, 124, 43 | -0.851 (0.5989) | -0.864 (0.5519) | -1.005 (0.6723)
  Week 36; n=64, 126, 43: number analyzed (Participants) | 64 | 126 | 43
  Week 36; n=64, 126, 43 | -0.916 (0.6141) | -0.927 (0.5400) | -0.917 (0.5504)
  Week 40; n=63, 126, 43: number analyzed (Participants) | 63 | 126 | 43
  Week 40; n=63, 126, 43 | -0.893 (0.6157) | -0.925 (0.5621) | -0.993 (0.6711)
  Week 44; n=63, 124, 43: number analyzed (Participants) | 63 | 124 | 43
  Week 44; n=63, 124, 43 | -0.800 (0.6764) | -0.905 (0.5289) | -0.970 (0.6065)
  Week 48; n=59, 121, 40: number analyzed (Participants) | 59 | 121 | 40
  Week 48; n=59, 121, 40 | -0.885 (0.6178) | -0.928 (0.5627) | -0.956 (0.5175)
  Week 52; n=64, 122, 41: number analyzed (Participants) | 64 | 122 | 41
  Week 52; n=64, 122, 41 | -0.947 (0.6918) | -0.938 (0.6125) | -1.004 (0.5527)
  Week 60; n=61, 120, 37: number analyzed (Participants) | 61 | 120 | 37
  Week 60; n=61, 120, 37 | -0.836 (0.6982) | -0.848 (0.6085) | -1.206 (0.5917)
  Week 64; n=62, 120, 36: number analyzed (Participants) | 62 | 120 | 36
  Week 64; n=62, 120, 36 | -0.876 (0.6971) | -0.943 (0.5711) | -1.095 (0.6365)
  Week 72; n=58, 110, 33: number analyzed (Participants) | 58 | 110 | 33
  Week 72; n=58, 110, 33 | -0.928 (0.6838) | -0.944 (0.5708) | -1.047 (0.6088)
  Week 80; n=57, 112, 37: number analyzed (Participants) | 57 | 112 | 37
  Week 80; n=57, 112, 37 | -0.949 (0.6909) | -0.954 (0.6221) | -1.138 (0.5574)
  Week 88; n=59, 109, 36: number analyzed (Participants) | 59 | 109 | 36
  Week 88; n=59, 109, 36 | -1.060 (0.6307) | -0.993 (0.5733) | -1.140 (0.5514)
  Week 96; n=54, 109, 35: number analyzed (Participants) | 54 | 109 | 35
  Week 96; n=54, 109, 35 | -1.016 (0.6093) | -0.994 (0.5669) | -1.214 (0.5580)
  Week 104; n=55, 114, 36: number analyzed (Participants) | 55 | 114 | 36
  Week 104; n=55, 114, 36 | -1.052 (0.5095) | -1.074 (0.5166) | -1.085 (0.5987)

19. Secondary Outcome: Percentage of Participants With Systemic Lupus International Collaborating Clinics (SLICC) -American College of Rheumatology (ACR) Damage Index Worsening Compared With Baseline at Week 52 and Week 104
Description: The SLICC-ACR Damage Index measures irreversible (not related to active inflammation) changes occurring since the diagnosis of SLE ascertained by clinical assessment and present for at least 6 months. The questionnaire contains 39 items covering 12 different organ systems which were scored on a numerical scale between 0 (no damage) to 7 (increasing disease damage). Individual ranges for organ systems were; ocular: 0-2, neuropsychiatric: 0-6, renal: 0-3, pulmonary: 0-5, cardiovascular:0-6, peripheral vascular: 0-5, gastrointestinal:0-5, musculoskeletal: 0-6, skin: 0-3, endocrine (diabetes): 0-1, gonadal:0-1 and malignancies: 0-2. The SLICC-ACR score was calculated by taking sum of the individual scores for 12 organ systems which ranges from 0 (no damage) to 45 (increasing disease damage) where higher score indicates increasing disease damage severity. Baseline value was the latest pre-dose assessment with a non-missing value, including those from unscheduled visits.
Time Frame: Baseline (Day 1), Week 52 and Week 104
Population: Modified Intent-to-Treat (MITT) Population
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Belimumab + Placebo | Belimumab + Rituximab | Belimumab + Standard Therapy
Number analyzed (Participants) | 72 | 144 | 47
Percentage of participants
  Week 52 | 1.4 [0 to 4.1] | 2.1 [0 to 4.4] | 2.1 [0 to 6.3]
  Week 104 | 5.6 [0.3 to 10.8] | 5.6 [1.8 to 9.3] | 6.4 [0 to 13.4]
Statistical Analysis 1: Comparison: Belimumab + Placebo vs Belimumab + Rituximab; Test type: Other; p = 0.7102, Regression, Logistic; Week 52; Odds Ratio (OR) = 1.55, 95% CI 2-sided [0.15 to 15.70] — Odds ratio at Week 52 was calculated using Logistic regression model with covariates:Baseline SLEDAI-2K,Baseline immunosuppressant,Baseline prednisone equivalent dose and treatment group. Belimumab+ Standard therapy arm was excluded from the model
Statistical Analysis 2: Comparison: Belimumab + Rituximab vs Belimumab + Standard Therapy; Test type: Other; Odds Ratio (OR) = 1.06, 95% CI 2-sided [0.10 to 10.71] — Odds ratio at Week 52 was calculated using Logistic regression model with covariates:Baseline SLEDAI-2K,Baseline immunosuppressant, Baseline prednisone equivalent dose and treatment group. Belimumab + Placebo arm was excluded from the model
Statistical Analysis 3: Comparison: Belimumab + Placebo vs Belimumab + Rituximab; Test type: Other; p = 0.8641, Regression, Logistic; Week 104; Odds Ratio (OR) = 0.90, 95% CI 2-sided [0.26 to 3.15] — Odds ratio at Week 104 was calculated using Logistic regression model with covariates:Baseline SLEDAI-2K,Baseline immunosuppressant,Baseline prednisone equivalent dose and treatment group. Belimumab + Standard therapy arm was excluded from the model
Statistical Analysis 4: Comparison: Belimumab + Rituximab vs Belimumab + Standard Therapy; Test type: Other; Odds Ratio (OR) = 1.22, 95% CI 2-sided [0.26 to 5.64] — Odds ratio at Week 104 was calculated using Logistic regression model with covariates:Baseline SLEDAI-2K,Baseline immunosuppressant,Baseline prednisone equivalent dose and treatment group. Belimumab + Placebo arm was excluded from the model

20. Secondary Outcome: Percentage of Participants That Met the Lupus Low Disease Activity State (LLDAS) Response Criteria by Visits (PI Assessed)
Description: Lupus low disease activity state (LLDAS) was defined as a state which, if sustained, was associated with a low likelihood of adverse outcome, considering disease activity and medication safety. The LLDAS response criteria were: (1) SLEDAI-2K <=4, with no activity in major organ systems (renal, CNS, cardiopulmonary, vasculitis, fever) and no hemolytic anemia or gastrointestinal activity; (2) no new features of lupus disease activity compared with the previous assessment; (3) PGA (scale 0-3), <=1; (4) current prednisolone (or equivalent) dose <=7.5 mg daily; and (5) well tolerated standard maintenance doses of immunosuppressive drugs and approved biological agents, excluding investigational drugs. Percentage of participants that met the LLDAS response criteria were reported.
Time Frame: Weeks 4, 8, 12, 16, 20, 24, 26, 28, 32, 36, 40, 44, 48, 52, 60, 64, 72, 80, 88, 96 and 104
Population: Modified Intent-to-Treat (MITT) Population
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Belimumab + Placebo | Belimumab + Rituximab | Belimumab + Standard Therapy
Number analyzed (Participants) | 72 | 144 | 47
Percentage of participants
  Week 4 | 0 [NA to NA] — NA indicates that data was not available as there was no participant who met the LLDAS response criteria. Hence, 95% CI could not be calculated. | 2.1 [0 to 4.4] | 2.1 [0 to 6.3]
  Week 8 | 9.7 [2.9 to 16.6] | 1.4 [0 to 3.3] | 10.6 [1.8 to 19.5]
  Week 12 | 8.3 [1.9 to 14.7] | 9.7 [4.9 to 14.6] | 6.4 [0 to 13.4]
  Week 16 | 11.1 [3.9 to 18.4] | 16.7 [10.6 to 22.8] | 19.1 [7.9 to 30.4]
  Week 20 | 11.1 [3.9 to 18.4] | 25.7 [18.6 to 32.8] | 19.1 [7.9 to 30.4]
  Week 24 | 12.5 [4.9 to 20.1] | 22.2 [15.4 to 29.0] | 36.2 [22.4 to 49.9]
  Week 26 | 22.2 [12.6 to 31.8] | 25.7 [18.6 to 32.8] | 34.0 [20.5 to 47.6]
  Week 28 | 20.8 [11.5 to 30.2] | 25.0 [17.9 to 32.1] | 34.0 [20.5 to 47.6]
  Week 32 | 29.2 [18.7 to 39.7] | 31.9 [24.3 to 39.6] | 36.2 [22.4 to 49.9]
  Week 36 | 30.6 [19.9 to 41.2] | 34.0 [26.3 to 41.8] | 29.8 [16.7 to 42.9]
  Week 40 | 22.2 [12.6 to 31.8] | 33.3 [25.6 to 41.0] | 38.3 [24.4 to 52.2]
  Week 44 | 30.6 [19.9 to 41.2] | 37.5 [29.6 to 45.4] | 31.9 [18.6 to 45.2]
  Week 48 | 26.4 [16.2 to 36.6] | 37.5 [29.6 to 45.4] | 31.9 [18.6 to 45.2]
  Week 52 | 27.8 [17.4 to 38.1] | 34.0 [26.3 to 41.8] | 29.8 [16.7 to 42.9]
  Week 60 | 26.4 [16.2 to 36.6] | 23.6 [16.7 to 30.5] | 36.2 [22.4 to 49.9]
  Week 64 | 20.8 [11.5 to 30.2] | 30.6 [23.0 to 38.1] | 31.9 [18.6 to 45.2]
  Week 72 | 22.2 [12.6 to 31.8] | 31.3 [23.7 to 38.8] | 31.9 [18.6 to 45.2]
  Week 80 | 18.1 [9.2 to 26.9] | 26.4 [19.2 to 33.6] | 34.0 [20.5 to 47.6]
  Week 88 | 23.6 [13.8 to 33.4] | 24.3 [17.3 to 31.3] | 29.8 [16.7 to 42.9]
  Week 96 | 20.8 [11.5 to 30.2] | 30.6 [23.0 to 38.1] | 36.2 [22.4 to 49.9]
  Week 104 | 20.8 [11.5 to 30.2] | 32.6 [25.0 to 40.3] | 38.3 [24.4 to 52.2]

21. Secondary Outcome: Percentage of Participants With a State of Disease Control Using the PI Assessment of SLEDAI-2K by Visit
Description: Percentage of participants with a state of disease control was defined as the percentage of participants with a SLEDAI-2K score <=2, achieved without immunosuppressants and with corticosteroids at a prednisone equivalent dose of <=5 mg/day, using the PI assessment of SLEDAI-2K. SLEDAI-2K consisted of 24 individual items within each of 9 organ systems. Each item was given a weighted score (1 to 8, higher score indicates increased activity) and summed if present at the time of visit or in preceding 10 days. SLEDAI-2K score was the sum of all 24 individual items from SLEDAI-2K, ranges from 0 (no symptoms) to 105 (presence of all defined symptoms), higher scores representing increased disease activity. Percentage of participants with a state of disease control using the PI assessment of SLEDAI-2K were summarized.
Time Frame: Weeks 4, 8, 12, 16, 20, 24, 26, 28, 32, 36, 40, 44, 48, 52, 60, 64, 72, 80, 88, 96, 104
Population: Modified Intent-to-Treat (MITT) Population
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Belimumab + Placebo | Belimumab + Rituximab | Belimumab + Standard Therapy
Number analyzed (Participants) | 72 | 144 | 47
Percentage of participants
  Week 4 | 2.8 [0 to 6.6] | 3.5 [0.5 to 6.5] | 8.5 [0.5 to 16.5]
  Week 8 | 13.9 [5.9 to 21.9] | 9.0 [4.3 to 13.7] | 21.3 [9.6 to 33.0]
  Week 12 | 11.1 [3.9 to 18.4] | 12.5 [7.1 to 17.9] | 19.1 [7.9 to 30.4]
  Week 16 | 15.3 [7.0 to 23.6] | 22.2 [15.4 to 29.0] | 29.8 [16.7 to 42.9]
  Week 20 | 13.9 [5.9 to 21.9] | 24.3 [17.3 to 31.3] | 31.9 [18.6 to 45.2]
  Week 24 | 18.1 [9.2 to 26.9] | 25.0 [17.9 to 32.1] | 34.0 [20.5 to 47.6]
  Week 26 | 15.3 [7.0 to 23.6] | 25.7 [18.6 to 32.8] | 25.5 [13.1 to 38.0]
  Week 28 | 11.1 [3.9 to 18.4] | 25.7 [18.6 to 32.8] | 36.2 [22.4 to 49.9]
  Week 32 | 15.3 [7.0 to 23.6] | 28.5 [21.1 to 35.8] | 31.9 [18.6 to 45.2]
  Week 36 | 19.4 [10.3 to 28.6] | 27.8 [20.5 to 35.1] | 27.7 [14.9 to 40.4]
  Week 40 | 16.7 [8.1 to 25.3] | 24.3 [17.3 to 31.3] | 23.4 [11.3 to 35.5]
  Week 44 | 18.1 [9.2 to 26.9] | 26.4 [19.2 to 33.6] | 27.7 [14.9 to 40.4]
  Week 48 | 18.1 [9.2 to 26.9] | 26.4 [19.2 to 33.6] | 27.7 [14.9 to 40.4]
  Week 52 | 19.4 [10.3 to 28.6] | 20.1 [13.6 to 26.7] | 27.7 [14.9 to 40.4]
  Week 60 | 18.1 [9.2 to 26.9] | 20.8 [14.2 to 27.5] | 23.4 [11.3 to 35.5]
  Week 64 | 11.1 [3.9 to 18.4] | 18.1 [11.8 to 24.3] | 27.7 [14.9 to 40.4]
  Week 72 | 9.7 [2.9 to 16.6] | 12.5 [7.1 to 17.9] | 23.4 [11.3 to 35.5]
  Week 80 | 8.3 [1.9 to 14.7] | 13.2 [7.7 to 18.7] | 31.9 [18.6 to 45.2]
  Week 88 | 11.1 [3.9 to 18.4] | 9.7 [4.9 to 14.6] | 21.3 [9.6 to 33.0]
  Week 96 | 8.3 [1.9 to 14.7] | 12.5 [7.1 to 17.9] | 31.9 [18.6 to 45.2]
  Week 104 | 8.3 [1.9 to 14.7] | 11.8 [6.5 to 17.1] | 23.4 [11.3 to 35.5]

22. Secondary Outcome: Percentage of Participants With a State of Clinical Remission Using the PI Assessment of SLEDAI-2K by Visit
Description: Percentage of participants with a state of clinical remission was defined as the percentage of participants with a clinical SLEDAI-2K score =0 (does not include anti-dsDNA and complement activity scores), achieved without immunosuppressants (which was allowed in Belimumab+ Standard therapy arm only) and with corticosteroids at a prednisone equivalent dose of 0 mg/day using the PI assessment of SLEDAI-2K. SLEDAI-2K consisted of 24 individual items within each of 9 organ systems. Each item was given a weighted score (1 to 8, higher score indicates increased activity) and summed if present at the time of visit or in preceding 10 days. The clinical SLEDAI-2K score was sum of 22 out of all 24 individual items from the SLEDAI-2K and ranges from 0 (no symptoms) to 101 (presence of all defined symptoms) with higher scores representing increased disease activity. Percentage of participants with a state of clinical remission using the PI assessment of SLEDAI-2K were summarized.
Time Frame: Weeks 60, 64, 72, 80, 88, 96 and 104
Population: Modified Intent-to-Treat (MITT) Population
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Belimumab + Placebo | Belimumab + Rituximab | Belimumab + Standard Therapy
Number analyzed (Participants) | 72 | 144 | 47
Percentage of participants
  Week 60 | 6.9 [1.1 to 12.8] | 3.5 [0.5 to 6.5] | 10.6 [1.8 to 19.5]
  Week 64 | 6.9 [1.1 to 12.8] | 5.6 [1.8 to 9.3] | 10.6 [1.8 to 19.5]
  Week 72 | 6.9 [1.1 to 12.8] | 3.5 [0.5 to 6.5] | 14.9 [4.7 to 25.1]
  Week 80 | 6.9 [1.1 to 12.8] | 4.2 [0.9 to 7.4] | 14.9 [4.7 to 25.1]
  Week 88 | 6.9 [1.1 to 12.8] | 2.1 [0 to 4.4] | 14.9 [4.7 to 25.1]
  Week 96 | 4.2 [0 to 8.8] | 4.2 [0.9 to 7.4] | 12.8 [3.2 to 22.3]
  Week 104 | 2.8 [0 to 6.6] | 3.5 [0.5 to 6.5] | 6.4 [0 to 13.4]

23. Secondary Outcome: Number of Participants With Serious Adverse Events (SAE) and Non-serious AE (Non-SAE)
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study treatment, whether or not considered related to the study treatment. A SAE is defined as any untoward medical occurrence that, at any dose results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent disability/incapacity, is a congenital anomaly/birth defect or any other situations as per medical or scientific judgment. Data for number of participants with SAE and non-SAE (>=5 %) has been summarized.
Time Frame: Up to Week 111 (including 8 weeks of safety follow-up)
Population: Intent-to-Treat Population comprised of all randomized participants who received at least one dose of study treatment (Belimumab or Rituximab or Placebo).
Measure: Count of Participants; unit: Participants
Arm/Group | Belimumab + Placebo | Belimumab + Rituximab | Belimumab + Standard Therapy
Number analyzed (Participants) | 72 | 144 | 76
Participants
  SAE | 10 | 32 | 15
  non-SAE | 48 | 109 | 53

24. Secondary Outcome: Number of Participants With Adverse Events of Special Interest (AESIs)
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study treatment, whether or not considered related to the study treatment. AESIs were Malignant Neoplasms, Post-Injection Systemic Reactions (PISR), All Infections of Special Interest (Opportunistic Infections (OI), Herpes Zoster (HZ), Tuberculosis (TB), and Sepsis), Depression (including mood disorders and anxiety)/suicide/self-injury and Deaths. Data for number of participants with AESIs has been summarized.
Time Frame: Up to Week 104
Population: Intent-to-Treat Population
Measure: Count of Participants; unit: Participants
Arm/Group | Belimumab + Placebo | Belimumab + Rituximab | Belimumab + Standard Therapy
Number analyzed (Participants) | 72 | 144 | 76
Participants
  Malignant Neoplasms | 1 | 1 | 1
  PISR | 7 | 19 | 4
  All Infections of Special Interest | 5 | 12 | 5
  Depression/suicide/self-injury | 9 | 16 | 5
  Deaths | 1 | 2 | 0

25. Secondary Outcome: Change From Baseline in Patient Global Assessment (PtGA) by Visits
Description: The Patient's Global Assessment (PtGA) of Disease Activity is a single-item, participant reported scale developed for the assessment of the participant's overall rating of their disease activity due to SLE. The scale measures disease activity ranging from 0 (Very Well) to 10 (Very Poor) and the higher score indicates severe disease activity. Baseline value was the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was defined as the post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1) and Weeks 8, 12, 26, 40, 52, 64, 72 and 104
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Belimumab + Placebo | Belimumab + Rituximab | Belimumab + Standard Therapy
Number analyzed (Participants) | 72 | 144 | 47
Scores on a scale
  Week 8; n=66, 132, 44: number analyzed (Participants) | 66 | 132 | 44
  Week 8; n=66, 132, 44 | -0.96 (2.751) | -1.06 (2.141) | -0.91 (2.848)
  Week 12; n=66, 133, 44: number analyzed (Participants) | 66 | 133 | 44
  Week 12; n=66, 133, 44 | -0.69 (2.237) | -1.07 (2.290) | -1.57 (2.756)
  Week 26; n=61, 115, 40: number analyzed (Participants) | 61 | 115 | 40
  Week 26; n=61, 115, 40 | -0.95 (2.765) | -1.50 (2.596) | -1.57 (2.450)
  Week 40; n=63, 123, 43: number analyzed (Participants) | 63 | 123 | 43
  Week 40; n=63, 123, 43 | -1.77 (2.624) | -1.60 (2.809) | -1.67 (2.962)
  Week 52; n=64, 120, 41: number analyzed (Participants) | 64 | 120 | 41
  Week 52; n=64, 120, 41 | -1.74 (2.752) | -1.82 (2.631) | -1.84 (3.228)
  Week 64; n=62, 117, 36: number analyzed (Participants) | 62 | 117 | 36
  Week 64; n=62, 117, 36 | -1.41 (2.985) | -1.96 (2.595) | -1.96 (3.034)
  Week 72; n=59, 107, 33: number analyzed (Participants) | 59 | 107 | 33
  Week 72; n=59, 107, 33 | -1.46 (3.209) | -1.81 (2.609) | -1.43 (3.487)
  Week 104; n=55, 111, 36: number analyzed (Participants) | 55 | 111 | 36
  Week 104; n=55, 111, 36 | -1.61 (2.589) | -2.00 (2.739) | -1.98 (2.895)

26. Secondary Outcome: Change From Baseline in Lupus Quality of Life (LupusQoL) Domain Scores by Visit
Description: LupusQoL is a SLE-specific health related qualify of life (HRQOL) instrument with 34 questions across 8 domains:Physical health(8 items),Pain(3 items),Planning(3 items),Intimate relationship(2 items),Burden to others(3 items),Emotional health(6 items),Body image(5 items),Fatigue(4 items). Questions were related to participants experience in prior 4 weeks.A 5-point Likert response format was used, ranging from 0(all of the time) to 4(never) for each question. Individual domain scores were reported which were calculated by taking sum of responses to all items within each domain. Individual domain scores range:Physical health(0-32),Pain(0-12),Planning(0-12),Intimate relationship(0-8),Burden to others(0-12),Emotional health(0-24),Body image(0-20),Fatigue(0-16). Higher score indicates better HRQOL. Baseline value was latest pre-dose assessment with a non-missing value including those from unscheduled visits. Change from Baseline was defined as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1) and Weeks 8, 12, 26, 40, 52, 64, 72 and 104
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Belimumab + Placebo | Belimumab + Rituximab | Belimumab + Standard Therapy
Number analyzed (Participants) | 72 | 144 | 47
Scores on a scale
  Physical health; Week 8; n=66, 132, 44: number analyzed (Participants) | 66 | 132 | 44
  Physical health; Week 8; n=66, 132, 44 | 3.0 (15.20) | 6.0 (15.08) | 6.3 (18.79)
  Physical health; Week 12; n=66, 133, 44: number analyzed (Participants) | 66 | 133 | 44
  Physical health; Week 12; n=66, 133, 44 | 3.5 (16.60) | 5.8 (17.15) | 6.4 (20.06)
  Physical health; Week 26; n=61, 115, 40: number analyzed (Participants) | 61 | 115 | 40
  Physical health; Week 26; n=61, 115, 40 | 3.3 (18.74) | 10.5 (17.27) | 11.6 (19.19)
  Physical health; Week 40; n=63, 122, 43: number analyzed (Participants) | 63 | 122 | 43
  Physical health; Week 40; n=63, 122, 43 | 8.5 (19.53) | 9.5 (19.29) | 8.2 (19.46)
  Physical health; Week 52; n=64, 120, 41: number analyzed (Participants) | 64 | 120 | 41
  Physical health; Week 52; n=64, 120, 41 | 8.1 (19.90) | 10.0 (20.16) | 11.6 (19.53)
  Physical health; Week 64; n=62, 117, 36: number analyzed (Participants) | 62 | 117 | 36
  Physical health; Week 64; n=62, 117, 36 | 5.8 (18.66) | 10.2 (18.60) | 9.5 (21.74)
  Physical health; Week 72; n=59, 107, 33: number analyzed (Participants) | 59 | 107 | 33
  Physical health; Week 72; n=59, 107, 33 | 7.0 (21.13) | 9.1 (18.84) | 8.5 (22.59)
  Physical health; Week 104; n=55, 111, 36: number analyzed (Participants) | 55 | 111 | 36
  Physical health; Week 104; n=55, 111, 36 | 6.2 (20.19) | 10.6 (19.96) | 7.2 (23.33)
  Pain; Week 8; n=66, 132, 44: number analyzed (Participants) | 66 | 132 | 44
  Pain; Week 8; n=66, 132, 44 | 5.8 (19.67) | 11.4 (18.55) | 10.4 (21.87)
  Pain; Week 12; n=66, 133, 44: number analyzed (Participants) | 66 | 133 | 44
  Pain; Week 12; n=66, 133, 44 | 7.5 (19.78) | 13.0 (20.81) | 6.1 (28.44)
  Pain; Week 26; n=61, 115, 40: number analyzed (Participants) | 61 | 115 | 40
  Pain; Week 26; n=61, 115, 40 | 7.0 (22.42) | 17.2 (21.54) | 13.1 (22.79)
  Pain; Week 40; n=63, 122, 43: number analyzed (Participants) | 63 | 122 | 43
  Pain; Week 40; n=63, 122, 43 | 12.3 (23.18) | 18.0 (22.70) | 12.6 (29.17)
  Pain; Week 52; n=64, 120, 41: number analyzed (Participants) | 64 | 120 | 41
  Pain; Week 52; n=64, 120, 41 | 13.9 (24.26) | 17.6 (23.62) | 15.7 (27.34)
  Pain; Week 64; n=62, 117, 36: number analyzed (Participants) | 62 | 117 | 36
  Pain; Week 64; n=62, 117, 36 | 10.2 (21.89) | 17.4 (23.59) | 13.2 (26.90)
  Pain; Week 72; n=59, 107, 33: number analyzed (Participants) | 59 | 107 | 33
  Pain; Week 72; n=59, 107, 33 | 13.1 (24.91) | 17.0 (22.66) | 11.9 (29.02)
  Pain; Week 104; n=55, 111, 36: number analyzed (Participants) | 55 | 111 | 36
  Pain; Week 104; n=55, 111, 36 | 13.8 (25.82) | 19.0 (22.59) | 12.5 (27.92)
  Planning; Week 8; n=66, 132, 44: number analyzed (Participants) | 66 | 132 | 44
  Planning; Week 8; n=66, 132, 44 | 3.4 (19.77) | 8.0 (18.21) | 10.0 (27.88)
  Planning; Week 12; n=66, 133, 44: number analyzed (Participants) | 66 | 133 | 44
  Planning; Week 12; n=66, 133, 44 | 4.5 (23.03) | 7.6 (20.15) | 7.8 (27.81)
  Planning; Week 26; n=61, 115, 40: number analyzed (Participants) | 61 | 115 | 40
  Planning; Week 26; n=61, 115, 40 | 3.4 (25.20) | 9.9 (21.28) | 12.1 (27.86)
  Planning; Week 40; n=63, 122, 43: number analyzed (Participants) | 63 | 122 | 43
  Planning; Week 40; n=63, 122, 43 | 11.6 (29.08) | 12.2 (22.30) | 10.7 (26.62)
  Planning; Week 52; n=64, 120, 41: number analyzed (Participants) | 64 | 120 | 41
  Planning; Week 52; n=64, 120, 41 | 11.6 (28.66) | 12.6 (23.89) | 14.0 (28.35)
  Planning; Week 64; n=62, 117, 36: number analyzed (Participants) | 62 | 117 | 36
  Planning; Week 64; n=62, 117, 36 | 7.8 (24.42) | 14.5 (23.65) | 7.2 (30.55)
  Planning; Week 72; n=59, 107, 33: number analyzed (Participants) | 59 | 107 | 33
  Planning; Week 72; n=59, 107, 33 | 9.2 (30.78) | 11.4 (20.97) | 6.6 (31.02)
  Planning; Week 104; n=55, 111, 36: number analyzed (Participants) | 55 | 111 | 36
  Planning; Week 104; n=55, 111, 36 | 12.1 (30.76) | 14.2 (20.77) | 8.8 (34.96)
  Intimate relationship; Week 8; n=51, 110, 36: number analyzed (Participants) | 51 | 110 | 36
  Intimate relationship; Week 8; n=51, 110, 36 | -1.2 (21.83) | 5.2 (20.63) | 7.6 (19.66)
  Intimate relationship; Week 12; n=52, 106, 36: number analyzed (Participants) | 52 | 106 | 36
  Intimate relationship; Week 12; n=52, 106, 36 | -2.6 (25.16) | 4.6 (23.42) | 7.6 (27.10)
  Intimate relationship; Week 26; n=48, 86, 30: number analyzed (Participants) | 48 | 86 | 30
  Intimate relationship; Week 26; n=48, 86, 30 | -1.3 (29.20) | 8.9 (24.32) | 14.2 (28.38)
  Intimate relationship; Week 40; n=50, 94, 30: number analyzed (Participants) | 50 | 94 | 30
  Intimate relationship; Week 40; n=50, 94, 30 | 4.3 (28.75) | 7.7 (25.01) | 15.8 (30.43)
  Intimate relationship; Week 52; n=51, 91, 30: number analyzed (Participants) | 51 | 91 | 30
  Intimate relationship; Week 52; n=51, 91, 30 | 4.7 (29.36) | 6.6 (22.54) | 15.8 (30.78)
  Intimate relationship; Week 64; n=47, 90, 25: number analyzed (Participants) | 47 | 90 | 25
  Intimate relationship; Week 64; n=47, 90, 25 | -4.5 (28.00) | 11.0 (25.41) | 12.5 (29.76)
  Intimate relationship; Week 72; n=42, 83, 21: number analyzed (Participants) | 42 | 83 | 21
  Intimate relationship; Week 72; n=42, 83, 21 | 0.0 (31.60) | 8.6 (23.82) | 5.4 (39.44)
  Intimate relationship; Week 104; n=40, 85,27: number analyzed (Participants) | 40 | 85 | 27
  Intimate relationship; Week 104; n=40, 85,27 | -0.3 (23.93) | 11.2 (25.59) | 4.6 (35.21)
  Burden to others; Week 8; n=66, 132, 44: number analyzed (Participants) | 66 | 132 | 44
  Burden to others; Week 8; n=66, 132, 44 | 7.3 (22.95) | 6.8 (20.56) | 10.6 (23.46)
  Burden to others; Week 12; n=66, 133, 44: number analyzed (Participants) | 66 | 133 | 44
  Burden to others; Week 12; n=66, 133, 44 | 11.4 (27.91) | 8.4 (23.65) | 6.4 (29.90)
  Burden to others; Week 26; n=61, 115, 40: number analyzed (Participants) | 61 | 115 | 40
  Burden to others; Week 26; n=61, 115, 40 | 8.7 (26.68) | 10.5 (27.42) | 7.5 (27.66)
  Burden to others; Week 40; n=63, 122, 43: number analyzed (Participants) | 63 | 122 | 43
  Burden to others; Week 40; n=63, 122, 43 | 13.9 (27.23) | 12.6 (26.94) | 12.0 (27.66)
  Burden to others; Week 52; n=64, 120, 41: number analyzed (Participants) | 64 | 120 | 41
  Burden to others; Week 52; n=64, 120, 41 | 16.5 (29.15) | 14.9 (27.03) | 15.0 (33.40)
  Burden to others; Week 64; n=62, 117, 36: number analyzed (Participants) | 62 | 117 | 36
  Burden to others; Week 64; n=62, 117, 36 | 14.4 (28.83) | 17.0 (26.67) | 12.3 (28.21)
  Burden to others; Week 72; n=59, 107, 33: number analyzed (Participants) | 59 | 107 | 33
  Burden to others; Week 72; n=59, 107, 33 | 17.1 (28.68) | 14.4 (28.77) | 11.1 (27.85)
  Burden to others; Week 104; n=55, 111, 36: number analyzed (Participants) | 55 | 111 | 36
  Burden to others; Week 104; n=55, 111, 36 | 18.9 (25.93) | 15.0 (29.25) | 12.7 (33.42)
  Emotional health; Week 8; n=66, 132, 44: number analyzed (Participants) | 66 | 132 | 44
  Emotional health; Week 8; n=66, 132, 44 | 5.2 (18.33) | 6.4 (16.87) | 11.6 (20.55)
  Emotional health; Week 12; n=66, 133, 44: number analyzed (Participants) | 66 | 133 | 44
  Emotional health; Week 12; n=66, 133, 44 | 8.1 (17.32) | 4.5 (19.67) | 9.1 (23.87)
  Emotional health; Week 26; n=61,115, 40: number analyzed (Participants) | 61 | 115 | 40
  Emotional health; Week 26; n=61,115, 40 | 7.7 (19.84) | 6.7 (17.35) | 10.1 (18.12)
  Emotional health; Week 40; n=63, 122, 43: number analyzed (Participants) | 63 | 122 | 43
  Emotional health; Week 40; n=63, 122, 43 | 9.7 (21.44) | 6.7 (20.85) | 9.4 (22.20)
  Emotional health; Week 52; n=64, 120, 41: number analyzed (Participants) | 64 | 120 | 41
  Emotional health; Week 52; n=64, 120, 41 | 10.2 (21.48) | 7.8 (20.63) | 11.4 (21.99)
  Emotional health; Week 64; n=62, 117, 36: number analyzed (Participants) | 62 | 117 | 36
  Emotional health; Week 64; n=62, 117, 36 | 8.1 (20.75) | 9.3 (20.73) | 8.1 (22.11)
  Emotional health; Week 72; n=59, 107, 33: number analyzed (Participants) | 59 | 107 | 33
  Emotional health; Week 72; n=59, 107, 33 | 8.8 (21.39) | 6.2 (19.05) | 6.6 (21.80)
  Emotional health; Week 104; n=55, 111, 36: number analyzed (Participants) | 55 | 111 | 36
  Emotional health; Week 104; n=55, 111, 36 | 6.8 (20.20) | 9.3 (19.67) | 10.5 (23.00)
  Body image; Week 8; n=60, 114, 37: number analyzed (Participants) | 60 | 114 | 37
  Body image; Week 8; n=60, 114, 37 | 5.7 (19.57) | 8.9 (19.26) | 5.7 (25.05)
  Body image; Week 12; n=58, 118, 39: number analyzed (Participants) | 58 | 118 | 39
  Body image; Week 12; n=58, 118, 39 | 1.9 (23.23) | 10.1 (20.73) | 5.9 (26.89)
  Body image; Week 26; n=56, 96, 33: number analyzed (Participants) | 56 | 96 | 33
  Body image; Week 26; n=56, 96, 33 | 5.8 (20.62) | 9.0 (25.03) | 5.7 (23.07)
  Body image; Week 40; n=54, 103, 35: number analyzed (Participants) | 54 | 103 | 35
  Body image; Week 40; n=54, 103, 35 | 8.9 (25.42) | 8.2 (24.82) | 5.1 (22.07)
  Body image; Week 52; n=55, 101, 33: number analyzed (Participants) | 55 | 101 | 33
  Body image; Week 52; n=55, 101, 33 | 7.9 (25.77) | 9.1 (24.07) | 10.3 (25.24)
  Body image; Week 64; n=52, 98, 27: number analyzed (Participants) | 52 | 98 | 27
  Body image; Week 64; n=52, 98, 27 | 6.0 (22.51) | 11.3 (23.08) | 7.7 (23.98)
  Body image; Week 72; n=44, 93, 25: number analyzed (Participants) | 44 | 93 | 25
  Body image; Week 72; n=44, 93, 25 | 7.8 (26.74) | 8.7 (24.91) | 2.5 (29.28)
  Body image; Week 104; n=48, 94, 28: number analyzed (Participants) | 48 | 94 | 28
  Body image; Week 104; n=48, 94, 28 | 4.4 (26.62) | 11.4 (25.65) | 3.5 (27.40)
  Fatigue; Week 8; n=66,132, 44: number analyzed (Participants) | 66 | 132 | 44
  Fatigue; Week 8; n=66,132, 44 | 9.8 (17.02) | 9.2 (18.40) | 8.5 (24.30)
  Fatigue; Week 12; n=66, 133, 44: number analyzed (Participants) | 66 | 133 | 44
  Fatigue; Week 12; n=66, 133, 44 | 8.2 (18.48) | 7.0 (17.96) | 10.4 (28.11)
  Fatigue; Week 26; n=61, 115, 40: number analyzed (Participants) | 61 | 115 | 40
  Fatigue; Week 26; n=61, 115, 40 | 8.6 (20.23) | 11.4 (20.12) | 11.9 (20.21)
  Fatigue; Week 40; n=63, 122, 43: number analyzed (Participants) | 63 | 122 | 43
  Fatigue; Week 40; n=63, 122, 43 | 11.9 (22.33) | 10.3 (22.41) | 11.3 (24.75)
  Fatigue; Week 52; n=64, 120, 41: number analyzed (Participants) | 64 | 120 | 41
  Fatigue; Week 52; n=64, 120, 41 | 14.2 (21.17) | 12.0 (20.95) | 16.6 (25.30)
  Fatigue; Week 64; n=62, 117, 36: number analyzed (Participants) | 62 | 117 | 36
  Fatigue; Week 64; n=62, 117, 36 | 10.5 (21.94) | 14.0 (20.35) | 10.8 (25.21)
  Fatigue; Week 72; n=59, 107, 33: number analyzed (Participants) | 59 | 107 | 33
  Fatigue; Week 72; n=59, 107, 33 | 12.1 (22.74) | 13.1 (18.31) | 11.6 (25.87)
  Fatigue; Week 104; n=55, 111, 36: number analyzed (Participants) | 55 | 111 | 36
  Fatigue; Week 104; n=55, 111, 36 | 9.4 (20.41) | 14.3 (20.18) | 9.7 (24.25)

27. Secondary Outcome: Change From Baseline in Functional Assessment of Chronic Illness Therapy (FACIT)-Fatigue Score by Visit
Description: The FACIT-Fatigue scale was a 13-item questionnaire completed by the participant, which provides a measure of fatigue/quality of life, with a 7-day recall period. The participant scored each item on a 5-point scale: 0 (Not at all) to 4 (Very much). The higher score for the questions, the greater the fatigue. The total score was the sum of the responses from all questions (inverted for reversed items) multiplied by 13, then divided by the number of questions answered, ranging from 0 (worse fatigue) to 52 (no fatigue) where a higher score indicates an improvement in the participant's health status and decrease in the score indicates worse fatigue/quality of life. Baseline value was the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was defined as the post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1) and Weeks 8, 12, 26, 40, 52, 64, 72 and 104
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Belimumab + Placebo | Belimumab + Rituximab | Belimumab + Standard Therapy
Number analyzed (Participants) | 72 | 144 | 47
Scores on a scale
  Week 8; n=66, 132, 44: number analyzed (Participants) | 66 | 132 | 44
  Week 8; n=66, 132, 44 | 4.2 (9.84) | 4.6 (8.84) | 4.8 (8.25)
  Week 12; n=66, 133, 44: number analyzed (Participants) | 66 | 133 | 44
  Week 12; n=66, 133, 44 | 4.7 (9.50) | 4.0 (9.86) | 3.8 (10.94)
  Week 26; n=61, 115, 40: number analyzed (Participants) | 61 | 115 | 40
  Week 26; n=61, 115, 40 | 3.1 (10.08) | 5.4 (9.17) | 4.1 (8.54)
  Week 40; n=63, 122, 43: number analyzed (Participants) | 63 | 122 | 43
  Week 40; n=63, 122, 43 | 6.0 (10.18) | 5.2 (10.80) | 5.2 (10.14)
  Week 52; n=64, 120, 41: number analyzed (Participants) | 64 | 120 | 41
  Week 52; n=64, 120, 41 | 6.5 (10.12) | 6.1 (10.84) | 5.1 (10.51)
  Week 64;n=62, 117, 36: number analyzed (Participants) | 62 | 117 | 36
  Week 64;n=62, 117, 36 | 4.9 (10.61) | 6.2 (9.72) | 4.6 (10.32)
  Week 72; n=59, 107, 33: number analyzed (Participants) | 59 | 107 | 33
  Week 72; n=59, 107, 33 | 5.6 (10.21) | 5.2 (10.31) | 2.9 (12.75)
  Week 104; n=55, 111, 36: number analyzed (Participants) | 55 | 111 | 36
  Week 104; n=55, 111, 36 | 5.7 (9.07) | 7.1 (11.50) | 3.1 (10.30)

28. Secondary Outcome: Percentage of Participants With Improvement in FACIT-Fatigue Score Exceeding the Minimal Clinically Important Difference (MCID, Greater Than or Equal to [>=]4)
Description: The FACIT-Fatigue scale was a 13-item questionnaire completed by the participant, which provides a measure of fatigue/quality of life, with a 7-day recall period. The participant scored each item on a 5-point scale: 0 (Not at all) to 4 (Very much). The larger the participant's response to the questions, the greater the fatigue. The total score was the sum of the responses (inverted for reversed items) multiplied by 13, then divided by the number of questions answered, ranging from 0 (worse fatigue) to 52 (no fatigue) where a higher score indicates an improvement in the participant's health status and decrease in the score indicates worse fatigue/quality of life. A participant was considered to had an improvement exceeding the minimal clinically important difference if they had >=4 points improvement in their FACIT-Fatigue Scale score from Baseline. Percentage of participants with improvement in FACIT-Fatigue scale score exceeding the MCID (>=4 points) were summarized.
Time Frame: Weeks 8, 12, 26, 40, 52, 64, 72 and 104
Population: as for outcome 15
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Belimumab + Placebo | Belimumab + Rituximab | Belimumab + Standard Therapy
Number analyzed (Participants) | 72 | 144 | 47
Percentage of participants
  Week 8; n=66, 132, 44: number analyzed (Participants) | 66 | 132 | 44
  Week 8; n=66, 132, 44 | 47.0 [34.9 to 59.0] | 51.5 [43.0 to 60.0] | 59.1 [44.6 to 73.6]
  Week 12; n=66, 133, 44: number analyzed (Participants) | 66 | 133 | 44
  Week 12; n=66, 133, 44 | 56.1 [44.1 to 68.0] | 50.4 [41.9 to 58.9] | 52.3 [37.5 to 67.0]
  Week 26; n=61, 115, 40: number analyzed (Participants) | 61 | 115 | 40
  Week 26; n=61, 115, 40 | 47.5 [35.0 to 60.1] | 56.5 [47.5 to 65.6] | 45.0 [29.6 to 60.4]
  Week 40; n=63, 122, 43: number analyzed (Participants) | 63 | 122 | 43
  Week 40; n=63, 122, 43 | 54.0 [41.7 to 66.3] | 54.1 [45.3 to 62.9] | 53.5 [38.6 to 68.4]
  Week 52; n=64, 120, 41: number analyzed (Participants) | 64 | 120 | 41
  Week 52; n=64, 120, 41 | 60.9 [49.0 to 72.9] | 58.3 [49.5 to 67.2] | 56.1 [40.9 to 71.3]
  Week 64; n=62, 117, 36: number analyzed (Participants) | 62 | 117 | 36
  Week 64; n=62, 117, 36 | 51.6 [39.2 to 64.1] | 59.8 [50.9 to 68.7] | 52.8 [36.5 to 69.1]
  Week 72; n=59, 107, 33: number analyzed (Participants) | 59 | 107 | 33
  Week 72; n=59, 107, 33 | 57.6 [45.0 to 70.2] | 57.0 [47.6 to 66.4] | 42.4 [25.6 to 59.3]
  Week 104; n=55, 111, 36: number analyzed (Participants) | 55 | 111 | 36
  Week 104; n=55, 111, 36 | 56.4 [43.3 to 69.5] | 62.2 [53.1 to 71.2] | 44.4 [28.2 to 60.7]

ADVERSE EVENTS:
Time Frame: All-cause mortality, serious adverse events (SAEs) and non-SAEs were collected up to Week 111 (including 8 weeks of safety follow-up).
Description: Intent-To-Treat (ITT) Population was used to assess the all-cause mortality, SAEs and non-SAEs which comprised of all randomized participants who received at least one dose of study treatment (Belimumab or Rituximab or placebo) .
Arm/Group | Belimumab + Placebo | Belimumab + Rituximab | Belimumab + Standard Therapy
All-Cause Mortality (participants affected / at risk) | 1/72 | 2/144 | 0/76
Serious Adverse Events (participants affected / at risk) | 10/72 | 32/144 | 15/76
Other Adverse Events (participants affected / at risk) | 48/72 | 109/144 | 53/76
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Belimumab + Placebo (N=72) | Belimumab + Rituximab (N=144) | Belimumab + Standard Therapy (N=76)
Chest pain (General disorders) | 1 (1) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Suicidal behaviour (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1)
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Vasculitis (Vascular disorders) | 0 (0) | 2 (3) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Abortion induced (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1)
Acute sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Adjustment disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Agranulocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Allergy to vaccine (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Angioedema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Arthritis bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Autoimmune hepatitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Bartholinitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Cervix carcinoma stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gangrene (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastritis viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Haematoma muscle (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Hemiparesis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Hepatitis A (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Hiatus hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperplasia of thymic epithelium (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Jugular vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Latent tuberculosis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Myocarditis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Nervous system disorder (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Neurogenic bladder (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Neuropsychiatric lupus (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Ocular myasthenia (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Orchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Pemphigoid (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pericarditis (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Pleuropericarditis (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Poisoning deliberate (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Post lumbar puncture syndrome (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1)
Respiratory tract infection viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Shrinking lung syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Spinal cord abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Sudden death (General disorders) | 0 (0) | 1 (1) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Suicide attempt (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Thrombophlebitis superficial (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Uterine haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Uterine polyp (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Vasculitis necrotising (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Volvulus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Belimumab + Placebo (N=72) | Belimumab + Rituximab (N=144) | Belimumab + Standard Therapy (N=76)
Headache (Nervous system disorders) | 13 (13) | 30 (44) | 8 (14)
Urinary tract infection (Infections and infestations) | 12 (16) | 23 (27) | 10 (27)
Nasopharyngitis (Infections and infestations) | 9 (13) | 23 (32) | 11 (18)
Upper respiratory tract infection (Infections and infestations) | 5 (6) | 22 (31) | 9 (12)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (5) | 12 (13) | 10 (13)
Bronchitis (Infections and infestations) | 6 (6) | 10 (10) | 7 (7)
Nausea (Gastrointestinal disorders) | 2 (3) | 18 (22) | 2 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 9 (9) | 4 (4)
Diarrhoea (Gastrointestinal disorders) | 6 (6) | 6 (6) | 5 (9)
Influenza (Infections and infestations) | 9 (12) | 4 (4) | 4 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (5) | 8 (8) | 4 (7)
Oral herpes (Infections and infestations) | 3 (6) | 9 (13) | 3 (7)
Vomiting (Gastrointestinal disorders) | 2 (2) | 11 (12) | 2 (4)
Pyrexia (General disorders) | 1 (1) | 10 (11) | 3 (9)
Abdominal pain upper (Gastrointestinal disorders) | 5 (7) | 7 (7) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 2 (2) | 7 (9) | 4 (4)
Sinusitis (Infections and infestations) | 4 (4) | 7 (8) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 9 (9) | 1 (1)
Depression (Psychiatric disorders) | 2 (2) | 6 (6) | 4 (4)
Hypertension (Vascular disorders) | 1 (1) | 7 (8) | 4 (5)
Chest pain (General disorders) | 1 (1) | 6 (8) | 4 (5)
Fatigue (General disorders) | 5 (7) | 5 (7) | 1 (2)
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 6 (9) | 3 (3) | 2 (2)
Pharyngitis (Infections and infestations) | 1 (1) | 4 (7) | 4 (4)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 4 (4) | 4 (4)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (3) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial

DOCUMENTS (2):
  • Study Protocol (2020-04-30): https://cdn.clinicaltrials.gov/large-docs/07/NCT03312907/Prot_000.pdf
  • Statistical Analysis Plan (2021-07-22): https://cdn.clinicaltrials.gov/large-docs/07/NCT03312907/SAP_001.pdf